CLINICAL TRIAL: NCT04742374
Title: Comparison of the Effects of 2 Therapeutic Plasmapheresis Techniques: Single Plasma Exchange and Double Filtration Plasmapheresis (DFPP) on Peripheral Lymphocyte Phenotypes in Patients With Chronic Inflammatory Demyelinating Polyradiculoneuropathy (CIDP). A Monocentric Prospective Study With a Single-Case Experimental Design
Brief Title: Effects of Single Plasma Exchange and Double Filtration Plasmapheresis (DFPP) on Peripheral Lymphocyte Phenotypes in Patients With Chronic Inflammatory Demyelinating Polyradiculoneuropathy
Acronym: LYMPHOARESIS
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: NIMAO/2020-01/OM001; 2020-A02879-30 (Other: ANSM)
Record Dates: First submitted 2021-01-26; First posted 2021-02-08 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-12

CONDITIONS: Polyradiculoneuropathy, Chronic Inflammatory Demyelinating
Keywords: Plasma exchange; Double filtration plasmapheresis
MeSH Terms: conditions — Polyradiculoneuropathy, Chronic Inflammatory Demyelinating | interventions — Blood Specimen Collection

STUDY DESIGN:
Intervention Model Description: Proof-of-concept, monocentric, prospective, Single-Case Experimental Design
Who Masked: Participant
Masking Description: Randomisation to one of two treatments before alternation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): Patients alternating single plasma exchange followed by double filtration plasmapheresis etc.
  Interventions: Biological: Blood sampling
- Group B (Experimental): Patients alternating double filtration plasmapheresis followed by single plasma exchange etc.
  Interventions: Biological: Blood sampling

INTERVENTIONS:
Biological: Blood sampling — Blood sampling before and after each type of cycle, Single Plasma Exchange or Double Filtration Plasmapheresis

SUMMARY:
CIDP, a rare disorder affecting young adults, causes gradual weakness of the limbs, areflexia and impaired sensory function. New CIDP phenotypes without antibodies but with modified cell profiles have been described. Treatments include corticotherapy, IVIg and plasmapheresis but the latter's action mechanisms remain unclear. Plasmapheresis supposedly removes toxic agents like antibodies from plasma but it is uncertain whether it has an immune-modulating effect. Also, the refining mechanisms of the two main plasmapheresis techniques - single plasma exchange and double filtration plasmapheresis (DFPP) - are different and unclear. This study aims to compare the evolution of peripheral lymphocyte profiles in patients with CIDP according to their treatment (single centrifugation plasmapheresis or DFPP) to better grasp the action mechanisms of both techniques.

ELIGIBILITY:
Inclusion Criteria:

* Patients with confirmed Chronic Inflammatory Demyelinating Polyneuropathy (CIDP) without pathogenic antibodies and stable under therapeutic plasmapheresis with one session every 2-3 weeks for at least two months.
* Patients who have given free written informed consent.
* Patients who have signed the consent form.
* Patients affiliated to or beneficiaries of a health insurance scheme.
* Adult patients (≥18 ans).
* Healthy subjects of the same age and sex

Exclusion Criteria:

* Patients Under the age of 18.
* Patients under immunosuppressive treatment for less than 3 months.
* Patients participating in Category 1 research involving human subjects.
* Patients in an exclusion period determined by another study.
* Patients under legal protection, guardianship or curatorship.
* Patients unable to express consent.
* Patients for whom it is impossible to give informed information.
* Pregnant, parturient or breastfeeding patients.
* Healthy subject with chronic pathology or drug treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2021-03-12 (Actual); Primary Completion 2023-12-18 (Actual); Study Completion 2023-12-18 (Actual)

PRIMARY OUTCOMES:
Cycle 1, Group A : TH1 cells BEFORE single plasma exchange | Day 0, Time 0
  5 mL of blood will be collected in an EDTA tube BEFORE single plasma exchange and the number of TH1 peripheral lymphocyte cells will be measured in %.
Cycle 1, Group A : TH1 cells AFTER single plasma exchange | Day 0, Hour 3
  5 mL of blood will be collected in an EDTA tube AFTER single plasma exchange and the number of TH1 peripheral lymphocyte cells will be measured in %.
Cycle 1, Group A : TH1 cells 7-10 days AFTER single plasma exchange | Day 7 -10
  5 mL of blood will be collected in an EDTA tube AFTER single plasma exchange and the number of TH1 peripheral lymphocyte cells will be measured in %.
Cycle 1, Group A : TH17 cells BEFORE first single plasma exchange | Day 0, Time 0
  5 mL of blood will be collected in an EDTA tube BEFORE single plasma exchange and the number of TH17 peripheral lymphocyte cells will be measured in %.
Cycle 1, Group A : TH17 cells AFTER single plasma exchange | Day 0, Hour 3
  5 mL of blood will be collected in an EDTA tube AFTER single plasma exchange and the number of TH17 peripheral lymphocyte cells will be measured in %.
Cycle 1, Group A : TH17 cells 7 - 10 days AFTER single plasma exchange | Day 7 - 10
  5 mL of blood will be collected in an EDTA tube AFTER single plasma exchange and the number of TH17 peripheral lymphocyte cells will be measured in %.
Cycle 1, Group A : T-reg cells BEFORE first single plasma exchange | Day 0, Hour 0
  5 mL of blood will be collected in an EDTA tube BEFORE single plasma exchange and the number of T-reg cells will be measured in %.
Cycle 1, Group A : T-reg cells AFTER single plasma exchange | Day 0, Hour 3
  5 mL of blood will be collected in an EDTA tube AFTER single plasma exchange and the number of T-reg cells will be measured in %.
Cycle 1, Group A : T-reg cells 7 - 10 days AFTER single plasma exchange | Day 7 - 10
  5 mL of blood will be collected in an EDTA tube AFTER single plasma exchange and the number of T-reg cells will be measured in %.
Cycle 1, Group B : TH1 cells BEFORE first double filtration plasmapheresis | Day 0, Hour 0
  5 mL of blood will be collected in an EDTA tube BEFORE double filtration plasmapheresis and the number of TH1 peripheral lymphocyte cells will be measured in %.
Cycle 1, Group B : TH1 cells AFTER the first double filtration plasmapheresis | Day 0, Hour 3
  5 mL of blood will be collected in an EDTA tube AFTER double filtration plasmapheresis and the number of TH1 peripheral lymphocyte cells will be measured in %.
Cycle 1, Group B : TH1 cells 7-10 days AFTER the first double filtration plasmapheresis | Day 7 - 10
  5 mL of blood will be collected in an EDTA tube AFTER double filtration plasmapheresis and the number of TH1 peripheral lymphocyte cells will be measured in %.
Cycle 1, Group B : TH17 cells BEFORE the first double filtration plasmapheresis | Day0, Hour 0
  5 mL of blood will be collected in an EDTA tube BEFORE double filtration plasmapheresis and the number of TH17 cells will be measured in %.
Cycle 1, Group B : TH17 cells AFTER the first double filtration plasmapheresis | Day 0, Hour 3
  5 mL of blood will be collected in an EDTA tube AFTER double filtration plasmapheresis and the number of TH17 cells will be measured in %.
Cycle 1, Group B : T17 cells 7-10 days AFTER double filtration plasmapheresis | Day 7-10
  5 mL of blood will be collected in an EDTA tube AFTER double filtration plasmapheresis and the number of TH17 cells will be measured in %.
Cycle 1, Group B : T-reg cells BEFORE double filtration plasmapheresis | Day 0, Hour 0
  5 mL of blood will be collected in an EDTA tube BEFORE double filtration plasmapheresis and the number of T-reg cells will be measured in %.
Cycle 1, Group B : T-reg cells AFTER double filtration plasmapheresis | Day 0, Hour 3
  5 mL of blood will be collected in an EDTA tube AFTER double filtration plasmapheresis and the number of T-reg cells will be measured in %.
Cycle 1, Group B : T-reg cells 7-10 days AFTER double filtration plasmapheresis | Day 7 - 10
  5 mL of blood will be collected in an EDTA tube AFTER double filtration plasmapheresis and the number of T-reg cells will be measured in %.
Cycle 2, Group A: TH1 cells BEFORE double filtration plasmapheresis | Day 0, Hour 0
  5 mL of blood will be collected in an EDTA tube BEFORE double filtration plasmapheresis and the number of TH1 cells will be measured in %.
Cycle 2, Group A: TH1 cells AFTER double filtration plasmapheresis | Day 0, Hour 3
  5 mL of blood will be collected in an EDTA tube AFTER double filtration plasmapheresis and the number of TH1 cells will be measured in %.
Cycle 2, Group A: TH1 cells 7-10 days AFTER double filtration plasmapheresis | Day 7 - 10
  5 mL of blood will be collected in an EDTA tube AFTER double filtration plasmapheresis and the number of TH1 cells will be measured in %.
Cycle 2, Group A: TH17 cells BEFORE double filtration plasmapheresis | Day 0, Hour 0
  5 mL of blood will be collected in an EDTA tube BEFORE double filtration plasmapheresis and the number of TH17 cells will be measured in %.
Cycle 2, Group A: TH17 cells AFTER double filtration plasmapheresis | Day 0, Hour 3
  5 mL of blood will be collected in an EDTA tube AFTER double filtration plasmapheresis and the number of TH17 cells will be measured in %.
Cycle 2, Group A: TH17 cells 7-10 days AFTER double filtration plasmapheresis | Day 7-10
  5 mL of blood will be collected in an EDTA tube AFTER double filtration plasmapheresis and the number of TH17 cells will be measured in %.
Cycle 2, Group A: T-reg cells BEFORE double filtration plasmapheresis | Day 0, Hour 0
  5 mL of blood will be collected in an EDTA tube BEFORE double filtration plasmapheresis and the number of T-reg cells will be measured in %.
Cycle 2, Group A: T-reg cells AFTER double filtration plasmapheresis | Day 0, Hour 3
  5 mL of blood will be collected in an EDTA tube AFTER double filtration plasmapheresis and the number of T-reg cells will be measured in %.
Cycle 2, Group A: T-reg cells 7-10 days AFTER double filtration plasmapheresis | Day 7-10
  5 mL of blood will be collected in an EDTA tube AFTER double filtration plasmapheresis and the number of T-reg cells will be measured in %.
Cycle 2, Group B: TH1 cells BEFORE single plasma exchange | Day 0, Hour 0
  5 mL of blood will be collected in an EDTA tube BEFORE single plasma exchange and the number of TH1 cells will be measured in %.
Cycle 2, Group B: TH1 cells AFTER single plasma exchange | Day 0, Hour 3
  5 mL of blood will be collected in an EDTA tube AFTER single plasma exchange and the number of TH1 cells will be measured in %.
Cycle 2, Group B: TH1 cells 7-10 days AFTER single plasma exchange | Day 7-10
  5 mL of blood will be collected in an EDTA tube AFTER single plasma exchange and the number of TH1 cells will be measured in %.
Cycle 2, Group B: T17 cells BEFORE single plasma exchange | Day 0, Hour 0
  5 mL of blood will be collected in an EDTA tube BEFORE single plasma exchange and the number of T17 cells will be measured in %.
Cycle 2, Group B: TH17 cells AFTER single plasma exchange | Day 0, Hour 3
  5 mL of blood will be collected in an EDTA tube AFTER single plasma exchange and the number of T17 cells will be measured in %.
Cycle 2, Group B: TH17 cells 7-10 days AFTER single plasma exchange | Day 7-10
  5 mL of blood will be collected in an EDTA tube AFTER single plasma exchange and the number of TH17 cells will be measured in %.
Cycle 2, Group B: T-reg cells BEFORE single plasma exchange | Day 0, Hour 0
  5 mL of blood will be collected in an EDTA tube BEFORE single plasma exchange and the number of T-reg cells will be measured in %.
Cycle 2, Group B: T-reg cells AFTER single plasma exchange | Day 0, Hour 3
  5 mL of blood will be collected in an EDTA tube AFTER single plasma exchange and the number of T-reg cells will be measured in %.
Cycle 2, Group B: T-reg cells 7-10 days AFTER single plasma exchange | Day 7-10
  5 mL of blood will be collected in an EDTA tube AFTER single plasma exchange and the number of T-reg cells will be measured in %.
Cycle 3, Group A: TH1 cells BEFORE single plasma exchange | Day 1, Hour 1
  5 mL of blood will be collected in an EDTA tube BEFORE single plasma exchange and the number of TH1 peripheral lymphocyte cells will be measured in %.
Cycle 3, Group A: TH1 cells AFTER single plasma exchange | Day 1, Hour 3
  5 mL of blood will be collected in an EDTA tube AFTER single plasma exchange and the number of TH1 peripheral lymphocyte cells will be measured in %.
Cycle 3, Group A: T1 cells 7-10 days AFTER single plasma exchange | Day 7 - 10
  5 mL of blood will be collected in an EDTA tube AFTER single plasma exchange and the number of TH1 peripheral lymphocyte cells will be measured in %.
Cycle 3, Group A: TH17 cells BEFORE single plasma exchange | Day 1, Hour 1
  5 mL of blood will be collected in an EDTA tube BEFORE single plasma exchange and the number of TH17 cells will be measured in %.
Cycle 3, Group A: TH17 cells AFTER single plasma exchange | Day 1, Hour 3
  5 mL of blood will be collected in an EDTA tube AFTER single plasma exchange and the number of TH17 cells will be measured in %.
Cycle 3, Group A: TH17 cells 7-10 days AFTER single plasma exchange | Day 7 - 10
  5 mL of blood will be collected in an EDTA tube AFTER single plasma exchange and the number of TH17 cells will be measured in %.
Cycle 3, Group A: T-reg cells BEFORE single plasma exchange | Day 0, Hour 0
  5 mL of blood will be collected in an EDTA tube BEFORE single plasma exchange and the number of T-reg cells will be measured in %.
Cycle 3, Group A: T-reg cells AFTER single plasma exchange | Day 0, Hour 3
  5 mL of blood will be collected in an EDTA tube AFTER single plasma exchange and the number of T-reg cells will be measured in %.
Cycle 3, Group A: T-reg cells 7-10 days AFTER single plasma exchange | Day 7-10
  5 mL of blood will be collected in an EDTA tube AFTER single plasma exchange and the number of T-reg cells will be measured in %.
Cycle 3, Group B: TH1 cells BEFORE double filtration plasmapheresis | Day 0, Hour 0
  5 mL of blood will be collected in an EDTA tube BEFORE double filtration plasmapheresis and the number of TH1 peripheral lymphocyte cells will be measured in %.
Cycle 3, Group B: TH1 cells AFTER double filtration plasmapheresis | Day 0, Hour 3
  5 mL of blood will be collected in an EDTA tube AFTER double filtration plasmapheresis and the number of TH1 peripheral lymphocyte cells will be measured in %.
Cycle 3, Group B: TH1 cells 7-10 days AFTER double filtration plasmapheresis | Day 7-10
  5 mL of blood will be collected in an EDTA tube AFTER double filtration plasmapheresis and the number of TH1 peripheral lymphocyte cells will be measured in %.
Cycle 3, Group B: TH17 cells BEFORE double filtration plasmapheresis | Day 0, Hour 0
  5 mL of blood will be collected in an EDTA tube BEFORE double filtration plasmapheresis and the number of TH17 cells will be measured in %.
Cycle 3, Group B: TH17 cells AFTER double filtration plasmapheresis | Day 0, Hour 3
  5 mL of blood will be collected in an EDTA tube AFTER double filtration plasmapheresis and the number of TH17 cells will be measured in %.
Cycle 3, Group B: TH17 cells 7-10 days AFTER double filtration plasmapheresis | Day 7-10
  5 mL of blood will be collected in an EDTA tube AFTER double filtration plasmapheresis and the number of TH17 cells will be measured in %.
Cycle 3, Group B: T-reg cells BEFORE double filtration plasmapheresis | Day 0, Hour 0
  5 mL of blood will be collected in an EDTA tube BEFORE double filtration plasmapheresis and the number of T-reg cells will be measured in %.
Cycle 3, Group B: T-reg cells AFTER double filtration plasmapheresis | Day 0, Hour 3
  5 mL of blood will be collected in an EDTA tube AFTER double filtration plasmapheresis and the number of T-reg cells will be measured in %.
Cycle 3, Group B: T-reg cells 7-10 days AFTER double filtration plasmapheresis | Day 7-10
  5 mL of blood will be collected in an EDTA tube AFTER double filtration plasmapheresis and the number of T-reg cells will be measured in %.
Cycle 4, Group A: T1 cells BEFORE double filtration plasmapheresis | Day 0, Hour 0
  5 mL of blood will be collected in an EDTA tube BEFORE double filtration plasmapheresis and the number of T1 peripheral lymphocyte cells will be measured in %.
Cycle 4, Group A: T1 cells AFTER double filtration plasmapheresis | Day 0, Hour 3
  5 mL of blood will be collected in an EDTA tube AFTER double filtration plasmapheresis and the number of T1 peripheral lymphocyte cells will be measured in %.
Cycle 4, Group A: TH1 cells 7-10 days AFTER double filtration plasmapheresis | Day 7 - 10
  5 mL of blood will be collected in an EDTA tube AFTER double filtration plasmapheresis and the number of TH1 peripheral lymphocyte cells will be measured in %.
Cycle 4, Group A: TH17 cells BEFORE double filtration plasmapheresis | Day 0, Hour 0
  5 mL of blood will be collected in an EDTA tube BEFORE double filtration plasmapheresis and the number of TH17 cells will be measured in %.
Cycle 4, Group A: TH17 cells AFTER double filtration plasmapheresis | Day 0, Hour 3
  5 mL of blood will be collected in an EDTA tube AFTER double filtration plasmapheresis and the number of TH17 cells will be measured in %.
Cycle 4, Group A: TH17 cells 7-10 days AFTER double filtration plasmapheresis | Day 7 - 10
  5 mL of blood will be collected in an EDTA tube AFTER double filtration plasmapheresis and the number of TH17 peripheral lymphocyte cells will be measured in %.
Cycle 4, Group A: T-reg cells BEFORE double filtration plasmapheresis | Day 0, Hour 0
  5 mL of blood will be collected in an EDTA tube BEFORE double filtration plasmapheresis and the number of T-reg cells will be measured in %.
Cycle 4, Group A: T-reg cells AFTER double filtration plasmapheresis | Day 0, Hour 3
  5 mL of blood will be collected in an EDTA tube AFTER double filtration plasmapheresis and the number of T-reg cells will be measured in %.
Cycle 4, Group A: T-reg cells 7-10 days AFTER double filtration plasmapheresis | Day 7 - 10
  5 mL of blood will be collected in an EDTA tube AFTER double filtration plasmapheresis and the number of T-reg peripheral lymphocyte cells will be measured in %.
Cycle 4, Group B : TH1 cells BEFORE single plasma exchange | Day 0, Hour 0
  5 mL of blood will be collected in an EDTA tube BEFORE single plasma exchange and the number of TH1 peripheral lymphocyte cells will be measured in %.
Cycle 4, Group B : TH1 cells AFTER single plasma exchange | Day 0, Hour 3
  5 mL of blood will be collected in an EDTA tube AFTER single plasma exchange and the number of TH1 peripheral lymphocyte cells will be measured in %.
Cycle 4, Group B : TH1 cells 7-10 days AFTER single plasma exchange | Day 7 -10
  5 mL of blood will be collected in an EDTA tube AFTER single plasma exchange and the number of TH1 peripheral lymphocyte cells will be measured in %.
Cycle 4, Group B : TH17 cells BEFORE single plasma exchange | Day 0, Hour 0
  5 mL of blood will be collected in an EDTA tube BEFORE single plasma exchange and the number of TH17 cells will be measured in %.
Cycle 4, Group B : TH17 cells AFTER single plasma exchange | Day 0, Hour 3
  5 mL of blood will be collected in an EDTA tube AFTER single plasma exchange and the number of TH17 cells will be measured in %.
Cycle 4, Group B : T17 cells 7-10 days AFTER single plasma exchange | Day 7 -10
  5 mL of blood will be collected in an EDTA tube AFTER single plasma exchange and the number of T1 peripheral lymphocyte cells will be measured in %.
Cycle 4, Group B : T-reg cells BEFORE single plasma exchange | Day 0, Hour 0
  5 mL of blood will be collected in an EDTA tube BEFORE single plasma exchange and the number of T-reg cells will be measured in %.
Cycle 4, Group B : T-reg cells AFTER single plasma exchange | Day 0, Hour 3
  5 mL of blood will be collected in an EDTA tube AFTER single plasma exchange and the number of T-reg cells will be measured in %.
Cycle 4, Group B : T-reg cells 7-10 days AFTER single plasma exchange | Day 7 - 10
  5 mL of blood will be collected in an EDTA tube AFTER single plasma exchange and the number of T-reg cells will be measured in %.
Cycle 5, Group A : TH1 cells BEFORE single plasma exchange | Day 0, Hour 0
  5 mL of blood will be collected in an EDTA tube BEFORE single plasma exchange and the number of TH1 peripheral lymphocyte cells will be measured in %.
Cycle 5, Group A : TH1 cells AFTER single plasma exchange | Day 0, Hour 3
  5 mL of blood will be collected in an EDTA tube AFTER single plasma exchange and the number of TH1 peripheral lymphocyte cells will be measured in %.
Cycle 5, Group A : TH1 cells 7-10 days AFTER single plasma exchange | Day 7 - 10
  5 mL of blood will be collected in an EDTA tube AFTER single plasma exchange and the number of TH1 cells will be measured in %.
Cycle 5, Group A : TH17 cells BEFORE single plasma exchange | Day 0, Hour 0
  5 mL of blood will be collected in an EDTA tube BEFORE single plasma exchange and the number of TH17 cells will be measured in %.
Cycle 5, Group A : TH17 cells AFTER single plasma exchange | Day 0, Hour 3
  5 mL of blood will be collected in an EDTA tube AFTER single plasma exchange and the number of TH17 cells will be measured in %.
Cycle 5, Group A : TH17 cells 7-10 days AFTER single plasma exchange | Day 7 - 10
  5 mL of blood will be collected in an EDTA tube AFTER single plasma exchange and the number of TH17 cells will be measured in %.
Cycle 5, Group A : T-reg cells BEFORE single plasma exchange | Day 0, Hour 0
  5 mL of blood will be collected in an EDTA tube BEFORE single plasma exchange and the number of T-reg cells will be measured in %.
Cycle 5, Group A : T-reg cells AFTER single plasma exchange | Day 0, Hour 3
  5 mL of blood will be collected in an EDTA tube AFTER single plasma exchange and the number of T-reg cells will be measured in %.
Cycle 5, Group A : T-reg cells 7-10 days AFTER single plasma exchange | Day 7 - 10
  5 mL of blood will be collected in an EDTA tube AFTER single plasma exchange and the number of T-reg cells will be measured in %.
Cycle 5, Group B : TH1 cells BEFORE double filtration plasmapheresis | Day 0, Hour 0
  5 mL of blood will be collected in an EDTA tube BEFORE double filtration plasmapheresis and the number of TH1 peripheral lymphocyte cells will be measured in %.
Cycle 5, Group B : TH1 cells AFTER double filtration plasmapheresis | Day 0, Hour 3
  5 mL of blood will be collected in an EDTA tube AFTER double filtration plasmapheresis and the number of TH1 peripheral lymphocyte cells will be measured in %.
Cycle 5, Group B : TH1 cells 7-10 days AFTER double filtration plasmapheresis | Day 7-10
  5 mL of blood will be collected in an EDTA tube AFTER double filtration plasmapheresis and the number of TH1 peripheral lymphocyte cells will be measured in %.
Cycle 5, Group B : TH17 cells BEFORE double filtration plasmapheresis | Day 0, Hour 0
  5 mL of blood will be collected in an EDTA tube BEFORE double filtration plasmapheresis and the number of TH17 cells will be measured in %.
Cycle 5, Group B : TH17 cells AFTER double filtration plasmapheresis | Day 0, Hour 3
  5 mL of blood will be collected in an EDTA tube AFTER double filtration plasmapheresis and the number of TH17 cells will be measured in %.
Cycle 5, Group B : TH17 cells 7-10 days AFTER double filtration plasmapheresis | Day 7-10
  5 mL of blood will be collected in an EDTA tube AFTER double filtration plasmapheresis and the number of TH17 cells will be measured in %.
Cycle 5, Group B : T-reg cells BEFORE double filtration plasmapheresis | Day 0, Hour 0
  5 mL of blood will be collected in an EDTA tube BEFORE double filtration plasmapheresis and the number of T-reg cells will be measured in %.
Cycle 5, Group B : T-reg cells AFTER double filtration plasmapheresis | Day 0, Hour 3
  5 mL of blood will be collected in an EDTA tube AFTER double filtration plasmapheresis and the number of T-reg cells will be measured in %.
Cycle 5, Group B : T-reg cells 7-10 days AFTER double filtration plasmapheresis | Day 7-10
  5 mL of blood will be collected in an EDTA tube AFTER double filtration plasmapheresis and the number of T-reg cells will be measured in %.
Cycle 6, Group A : TH1 cells BEFORE double filtration plasmapheresis | Day 0 Hour 0
  5 mL of blood will be collected in an EDTA tube BEFORE double filtration plasmapheresis and the number of TH1 peripheral lymphocyte cells will be measured in %.
Cycle 6, Group A : TH1 cells AFTER double filtration plasmapheresis | Day 0 Hour 3
  5 mL of blood will be collected in an EDTA tube AFTER double filtration plasmapheresis and the number of TH1 peripheral lymphocyte cells will be measured in %.
Cycle 6, Group A : TH1 cells 7-10 days AFTER double filtration plasmapheresis | Day 7-10
  5 mL of blood will be collected in an EDTA tube 7-10 days AFTER double filtration plasmapheresis and the number of TH1 peripheral lymphocyte cells will be measured in %.
Cycle 6, Group A : TH17 cells BEFORE double filtration plasmapheresis | Day 0 Hour 0
  5 mL of blood will be collected in an EDTA tube BEFORE double filtration plasmapheresis and the number of TH17 cells will be measured in %.
Cycle 6, Group A : TH17 cells AFTER double filtration plasmapheresis | Day 0 Hour 3
  5 mL of blood will be collected in an EDTA tube AFTER double filtration plasmapheresis and the number of TH17 cells will be measured in %.
Cycle 6, Group A : TH17 cells 7-10 days AFTER double filtration plasmapheresis | Day 7-10
  5 mL of blood will be collected in an EDTA tube 7-10 days AFTER double filtration plasmapheresis and the number of TH17 cells will be measured in %.
Cycle 6, Group A : T-reg cells BEFORE double filtration plasmapheresis | Day 0 Hour 0
  5 mL of blood will be collected in an EDTA tube BEFORE double filtration plasmapheresis and the number of T-reg cells will be measured in %.
Cycle 6, Group A : T-reg cells AFTER double filtration plasmapheresis | Day 0 Hour 3
  5 mL of blood will be collected in an EDTA tube AFTER double filtration plasmapheresis and the number of T-reg cells will be measured in %.
Cycle 6, Group A : T-reg cells 7-10 days AFTER double filtration plasmapheresis | Day 7-10
  5 mL of blood will be collected in an EDTA tube 7-10 days AFTER double filtration plasmapheresis and the number of T-reg cells will be measured in %.
Cycle 6, Group B : TH1 cells BEFORE single plasma exchange | Day 0 Hour 0
  5 mL of blood will be collected in an EDTA tube BEFORE single plasma exchange and the number of TH1 peripheral lymphocyte cells will be measured in %.
Cycle 6, Group B : TH1 cells AFTER single plasma exchange | Day 0 Hour 3
  5 mL of blood will be collected in an EDTA tube AFTER single plasma exchange and the number of TH1 peripheral lymphocyte cells will be measured in %.
Cycle 6, Group B : TH1 cells 7-10 days AFTER single plasma exchange | Day 7-10
  5 mL of blood will be collected in an EDTA tube AFTER single plasma exchange and the number of TH1 peripheral lymphocyte cells will be measured in %.
Cycle 6, Group B : TH17 cells BEFORE single plasma exchange | Day 0 Hour 0
  5 mL of blood will be collected in an EDTA tube BEFORE single plasma exchange and the number of TH17 cells will be measured in %.
Cycle 6, Group B : TH17 cells AFTER single plasma exchange | Day 0 Hour 3
  5 mL of blood will be collected in an EDTA tube AFTER single plasma exchange and the number of TH17 cells will be measured in %.
Cycle 6, Group B : TH17 cells 7-10 days AFTER single plasma exchange | Day 7-10
  5 mL of blood will be collected in an EDTA tube AFTER single plasma exchange and the number of TH17 cells will be measured in %.
Cycle 6, Group B : T-reg cells BEFORE single plasma exchange | Day 0 Hour 0
  5 mL of blood will be collected in an EDTA tube BEFORE single plasma exchange and the number of T-reg cells will be measured in %.
Cycle 6, Group B : T-reg cells AFTER single plasma exchange | Day 0 Hour 3
  5 mL of blood will be collected in an EDTA tube AFTER single plasma exchange and the number of T-reg cells will be measured in %.
Cycle 6, Group B : T-reg cells 7-10 days AFTER single plasma exchange | Day 7-10
  5 mL of blood will be collected in an EDTA tube AFTER single plasma exchange and the number of T-reg cells will be measured in %.

SECONDARY OUTCOMES:
Cycle 1, Group A : T4 lymphocytes BEFORE single plasma exchange | Day 0 Hour 0
  5 mL of blood will be collected in an EDTA tube BEFORE single plasma exchange and cell counts will be made by flow cytometry after marking with specific fluorescent antibodies (Luminex) and measured as a percentage.
Cycle 1, Group A : T4-DR+ lymphocytes BEFORE single plasma exchange | Day 0 Hour 0
  5 mL of blood will be collected in an EDTA tube BEFORE single plasma exchange and cell counts will be made by flow cytometry after marking with specific fluorescent antibodies (Luminex) and measured as a percentage.
Cycle 1, Group A : T8 lymphocytes BEFORE single plasma exchange | Day 0 Hour 0
  5 mL of blood will be collected in an EDTA tube BEFORE single plasma exchange and cell counts will be made by flow cytometry after marking with specific fluorescent antibodies (Luminex) and measured as a percentage.
Cycle 1, Group A : T8 DR+ lymphocytes BEFORE single plasma exchange | Day 0 Hour 0
  5 mL of blood will be collected in an EDTA tube BEFORE single plasma exchange and cell counts will be made by flow cytometry after marking with specific fluorescent antibodies (Luminex) and measured as a percentage.
Cycle 1, Group A : B lymphocytes BEFORE single plasma exchange | Day 0 Hour 0
  5 mL of blood will be collected in an EDTA tube BEFORE single plasma exchange and cell counts will be made by flow cytometry after marking with specific fluorescent antibodies (Luminex) and measured as a percentage.
Cycle 1, Group A : CD45RA+CCR7+ cells BEFORE single plasma exchange | Day 0 Hour 0
  5 mL of blood will be collected in an EDTA tube BEFORE single plasma exchange and cell counts will be made by flow cytometry after marking with specific fluorescent antibodies (Luminex) and measured as a percentage.
Cycle 1, Group A : CD45RA-CCR7+ cells BEFORE single plasma exchange | Day 0 Hour 0
  5 mL of blood will be collected in an EDTA tube BEFORE single plasma exchange and cell counts will be made by flow cytometry after marking with specific fluorescent antibodies (Luminex) and measured as a percentage.
Cycle 1, Group A : CD45RA-CCR7- cells BEFORE single plasma exchange | Day 0 Hour 0
  5 mL of blood will be collected in an EDTA tube BEFORE single plasma exchange and cell counts will be made by flow cytometry after marking with specific fluorescent antibodies (Luminex) and measured as a percentage.
Cycle 1, Group A : CCR6-CXCR3- cells BEFORE single plasma exchange | Day 0 Hour 0
  5 mL of blood will be collected in an EDTA tube BEFORE single plasma exchange and cell counts will be made by flow cytometry after marking with specific fluorescent antibodies (Luminex) and measured as a percentage.
Cycle 1, Group A : T4 lymphocytes AFTER single plasma exchange | Day 0 Hour 3
  5 mL of blood will be collected in an EDTA tube AFTER single plasma exchange and cell counts will be made by flow cytometry after marking with specific fluorescent antibodies (Luminex) and measured as a percentage.
Cycle 1, Group A : T4-DR+ lymphocytes AFTER single plasma exchange | Day 0 Hour 3
  5 mL of blood will be collected in an EDTA tube AFTER single plasma exchange and cell counts will be made by flow cytometry after marking with specific fluorescent antibodies (Luminex) and measured as a percentage.
Cycle 1, Group A : T8 lymphocytes AFTER single plasma exchange | Day 0 Hour 3
  5 mL of blood will be collected in an EDTA tube AFTER single plasma exchange and cell counts will be made by flow cytometry after marking with specific fluorescent antibodies (Luminex) and measured as a percentage.
Cycle 1, Group A : T8 DR+ lymphocytes AFTER single plasma exchange | Day 0 Hour 3
  5 mL of blood will be collected in an EDTA tube AFTER single plasma exchange and cell counts will be made by flow cytometry after marking with specific fluorescent antibodies (Luminex) and measured as a percentage.
Cycle 1, Group A : B lymphocytes AFTER single plasma exchange | Day 0 Hour 3
  5 mL of blood will be collected in an EDTA tube AFTER single plasma exchange and cell counts will be made by flow cytometry after marking with specific fluorescent antibodies (Luminex) and measured as a percentage.
Cycle 1, Group A : CD45RA+CCR7+ cells AFTER single plasma exchange | Day 0 Hour 3
  5 mL of blood will be collected in an EDTA tube AFTER single plasma exchange and cell counts will be made by flow cytometry after marking with specific fluorescent antibodies (Luminex) and measured as a percentage.
Cycle 1, Group A : CD45RA-CCR7+ cells AFTER single plasma exchange | Day 0 Hour 3
  5 mL of blood will be collected in an EDTA tube AFTER single plasma exchange and cell counts will be made by flow cytometry after marking with specific fluorescent antibodies (Luminex) and measured as a percentage.
Cycle 1, Group A : CD45RA-CCR7- cells AFTER single plasma exchange | Day 0 Hour 3
  5 mL of blood will be collected in an EDTA tube AFTER single plasma exchange and cell counts will be made by flow cytometry after marking with specific fluorescent antibodies (Luminex) and measured as a percentage.
Cycle 1, Group A : CR6-CXCR3- cells AFTER single plasma exchange | Day 0 Hour 3
  5 mL of blood will be collected in an EDTA tube AFTER single plasma exchange and cell counts will be made by flow cytometry after marking with specific fluorescent antibodies (Luminex) and measured as a percentage.
Cycle 1, Group A : T4 lymphocytes 7-10 days AFTER single plasma exchange | Day 7-10
  5 mL of blood will be collected in an EDTA tube AFTER single plasma exchange and cell counts will be made by flow cytometry after marking with specific fluorescent antibodies (Luminex) and measured as a percentage.
Cycle 1, Group A : T4-DR+ lymphocytes 7-10 days AFTER single plasma exchange | Day 7-10
  5 mL of blood will be collected in an EDTA tube AFTER single plasma exchange and cell counts will be made by flow cytometry after marking with specific fluorescent antibodies (Luminex) and measured as a percentage.
Cycle 1, Group A : T8 lymphocytes 7-10 days AFTER single plasma exchange | Day 7-10
  5 mL of blood will be collected in an EDTA tube AFTER single plasma exchange and cell counts will be made by flow cytometry after marking with specific fluorescent antibodies (Luminex) and measured as a percentage.
Cycle 1, Group A : T8 DR+ lymphocytes 7-10 days AFTER single plasma exchange | Day 7-10
  5 mL of blood will be collected in an EDTA tube AFTER single plasma exchange and cell counts will be made by flow cytometry after marking with specific fluorescent antibodies (Luminex) and measured as a percentage.
Cycle 1, Group A : B lymphocytes 7-10 days AFTER single plasma exchange | Day 7-10
  5 mL of blood will be collected in an EDTA tube AFTER single plasma exchange and cell counts will be made by flow cytometry after marking with specific fluorescent antibodies (Luminex) and measured as a percentage.
Cycle 1, Group A : CD45RA+CCR7+ cells 7-10 days AFTER single plasma exchange | Day 7-10
  5 mL of blood will be collected in an EDTA tube AFTER single plasma exchange and cell counts will be made by flow cytometry after marking with specific fluorescent antibodies (Luminex) and measured as a percentage.
Cycle 1, Group A : CD45RA-CCR7+ cells 7-10 days AFTER single plasma exchange | Day 7-10
  5 mL of blood will be collected in an EDTA tube AFTER single plasma exchange and cell counts will be made by flow cytometry after marking with specific fluorescent antibodies (Luminex) and measured as a percentage.
Cycle 1, Group A : CD45RA-CCR7- cells 7-10 days AFTER single plasma exchange | Day 7-10
  5 mL of blood will be collected in an EDTA tube AFTER single plasma exchange and cell counts will be made by flow cytometry after marking with specific fluorescent antibodies (Luminex) and measured as a percentage.
Cycle 1, Group A : CCR6-CXCR3- cells 7-10 days AFTER single plasma exchange | Day 7-10
  5 mL of blood will be collected in an EDTA tube AFTER single plasma exchange and cell counts will be made by flow cytometry after marking with specific fluorescent antibodies (Luminex) and measured as a percentage.
Cycle 1, Group B: T4 lymphocytes BEFORE double filtration plasmapheresis | Day 0 Hour 0
  5 mL of blood will be collected in an EDTA tube BEFORE double filtration plasmapheresis and cell counts will be made by flow cytometry after marking with specific fluorescent antibodies (Luminex) and measured as a percentage.
Cycle 1, Group B: T4 DR+ lymphocytes BEFORE double filtration plasmapheresis | Day 0 Hour 0
  5 mL of blood will be collected in an EDTA tube BEFORE double filtration plasmapheresis and cell counts will be made by flow cytometry after marking with specific fluorescent antibodies (Luminex) and measured as a percentage.
Cycle 1, Group B: T8 lymphocytes BEFORE double filtration plasmapheresis | Day 0 Hour 0
  5 mL of blood will be collected in an EDTA tube BEFORE double filtration plasmapheresis and cell counts will be made by flow cytometry after marking with specific fluorescent antibodies (Luminex) and measured as a percentage.
Cycle 1, Group B: T8 DR+ lymphocytes BEFORE double filtration plasmapheresis | Day 0 Hour 0
  5 mL of blood will be collected in an EDTA tube BEFORE double filtration plasmapheresis and cell counts will be made by flow cytometry after marking with specific fluorescent antibodies (Luminex) and measured as a percentage.
Cycle 1, Group B: B lymphocytes BEFORE double filtration plasmapheresis | Day 0 Hour 0
  5 mL of blood will be collected in an EDTA tube BEFORE double filtration plasmapheresis and cell counts will be made by flow cytometry after marking with specific fluorescent antibodies (Luminex) and measured as a percentage.
Cycle 1, Group B: CD45RA+CCR7+ cells BEFORE double filtration plasmapheresis | Day 0 Hour 0
  5 mL of blood will be collected in an EDTA tube BEFORE double filtration plasmapheresis and cell counts will be made by flow cytometry after marking with specific fluorescent antibodies (Luminex) and measured as a percentage.
Cycle 1, Group B: CD45RA-CCR7+ cells BEFORE double filtration plasmapheresis | Day 0 Hour 0
  5 mL of blood will be collected in an EDTA tube BEFORE double filtration plasmapheresis and cell counts will be made by flow cytometry after marking with specific fluorescent antibodies (Luminex) and measured as a percentage.
Cycle 1, Group B: CD45RA-CCR7- cells BEFORE double filtration plasmapheresis | Day 0 Hour 0
  5 mL of blood will be collected in an EDTA tube BEFORE double filtration plasmapheresis and cell counts will be made by flow cytometry after marking with specific fluorescent antibodies (Luminex) and measured as a percentage.
Cycle 1, Group B: CCR6-CXCR3- cells BEFORE double filtration plasmapheresis | Day 0 Hour 0
  5 mL of blood will be collected in an EDTA tube BEFORE double filtration plasmapheresis and cell counts will be made by flow cytometry after marking with specific fluorescent antibodies (Luminex) and measured as a percentage.
Cycle 1, Group B:T4 lymphocytes AFTER double filtration plasmapheresis | Day 0 Hour 3
  5 mL of blood will be collected in an EDTA tube AFTER double filtration plasmapheresis and cell counts will be made by flow cytometry after marking with specific fluorescent antibodies (Luminex) and measured as a percentage.
Cycle 1, Group B:T4 DR+ lymphocytes AFTER double filtration plasmapheresis | Day 0 Hour 3
  5 mL of blood will be collected in an EDTA tube AFTER double filtration plasmapheresis and cell counts will be made by flow cytometry after marking with specific fluorescent antibodies (Luminex) and measured as a percentage.
Cycle 1, Group B:T8 lymphocytes AFTER double filtration plasmapheresis | Day 0 Hour 3
  5 mL of blood will be collected in an EDTA tube AFTER double filtration plasmapheresis and cell counts will be made by flow cytometry after marking with specific fluorescent antibodies (Luminex) and measured as a percentage.
Cycle 1, Group B:T8 DR+ lymphocytes AFTER double filtration plasmapheresis | Day 0 Hour 3
  5 mL of blood will be collected in an EDTA tube AFTER double filtration plasmapheresis and cell counts will be made by flow cytometry after marking with specific fluorescent antibodies (Luminex) and measured as a percentage.
Cycle 1, Group B: B lymphocytes AFTER double filtration plasmapheresis | Day 0 Hour 3
  5 mL of blood will be collected in an EDTA tube AFTER double filtration plasmapheresis and cell counts will be made by flow cytometry after marking with specific fluorescent antibodies (Luminex) and measured as a percentage.
Cycle 1, Group B: CD45RA+CCR7+ cells AFTER double filtration plasmapheresis | Day 0 Hour 3
  5 mL of blood will be collected in an EDTA tube AFTER double filtration plasmapheresis and cell counts will be made by flow cytometry after marking with specific fluorescent antibodies (Luminex) and measured as a percentage.
Cycle 1, Group B: CD45RA-CCR7+ cells AFTER double filtration plasmapheresis | Day 0 Hour 3
  5 mL of blood will be collected in an EDTA tube AFTER double filtration plasmapheresis and cell counts will be made by flow cytometry after marking with specific fluorescent antibodies (Luminex) and measured as a percentage.
Cycle 1, Group B: CD45RA-CCR7- cells AFTER double filtration plasmapheresis | Day 0 Hour 3
  5 mL of blood will be collected in an EDTA tube AFTER double filtration plasmapheresis and cell counts will be made by flow cytometry after marking with specific fluorescent antibodies (Luminex) and measured as a percentage.
Cycle 1, Group B: CCR6-CXCR3- cells AFTER double filtration plasmapheresis | Day 0 Hour 3
  5 mL of blood will be collected in an EDTA tube AFTER double filtration plasmapheresis and cell counts will be made by flow cytometry after marking with specific fluorescent antibodies (Luminex) and measured as a percentage.
Cycle 1, Group B: T4 lymphocytes 7-10 days AFTER double filtration plasmapheresis | Day 7-10
  5 mL of blood will be collected in an EDTA tube 7-10 days AFTER double filtration plasmapheresis and cell counts will be made by flow cytometry after marking with specific fluorescent antibodies (Luminex) and measured as a percentage.
Cycle 1, Group B: T4 DR+ lymphocytes 7-10 days AFTER double filtration plasmapheresis | Day 7-10
  5 mL of blood will be collected in an EDTA tube 7-10 days AFTER double filtration plasmapheresis and cell counts will be made by flow cytometry after marking with specific fluorescent antibodies (Luminex) and measured as a percentage.
Cycle 1, Group B: T8 lymphocytes 7-10 days AFTER double filtration plasmapheresis | Day 7-10
  5 mL of blood will be collected in an EDTA tube 7-10 days AFTER double filtration plasmapheresis and cell counts will be made by flow cytometry after marking with specific fluorescent antibodies (Luminex) and measured as a percentage.
Cycle 1, Group B: T8 DR+ lymphocytes 7-10 days AFTER double filtration plasmapheresis | Day 7-10
  5 mL of blood will be collected in an EDTA tube 7-10 days AFTER double filtration plasmapheresis and cell counts will be made by flow cytometry after marking with specific fluorescent antibodies (Luminex) and measured as a percentage.
Cycle 1, Group B: B lymphocytes 7-10 days AFTER double filtration plasmapheresis | Day 7-10
  5 mL of blood will be collected in an EDTA tube 7-10 days AFTER double filtration plasmapheresis and cell counts will be made by flow cytometry after marking with specific fluorescent antibodies (Luminex) and measured as a percentage.
Cycle 1, Group B: CD45RA+CCR7+ cells 7-10 days AFTER double filtration plasmapheresis | Day 7-10
  5 mL of blood will be collected in an EDTA tube 7-10 days AFTER double filtration plasmapheresis and cell counts will be made by flow cytometry after marking with specific fluorescent antibodies (Luminex) and measured as a percentage.
Cycle 1, Group B: CD45RA-CCR7+ cells 7-10 days AFTER double filtration plasmapheresis | Day 7-10
  5 mL of blood will be collected in an EDTA tube 7-10 days AFTER double filtration plasmapheresis and cell counts will be made by flow cytometry after marking with specific fluorescent antibodies (Luminex) and measured as a percentage.
Cycle 1, Group B: CD45RA-CCR7- cells 7-10 days AFTER double filtration plasmapheresis | Day 7-10
  5 mL of blood will be collected in an EDTA tube 7-10 days AFTER double filtration plasmapheresis and cell counts will be made by flow cytometry after marking with specific fluorescent antibodies (Luminex) and measured as a percentage.
Cycle 1, Group B: CCR6-CXCR3- cells 7-10 days AFTER double filtration plasmapheresis | Day 7-10
  5 mL of blood will be collected in an EDTA tube 7-10 days AFTER double filtration plasmapheresis and cell counts will be made by flow cytometry after marking with specific fluorescent antibodies (Luminex) and measured as a percentage.
Cycle 2, Group A : T4 lymphocytes BEFORE double filtration plasmapheresis | Day 0 Hour 0
  5 mL of blood will be collected in an EDTA tube BEFORE double filtration plasmapheresis and cell counts will be made by flow cytometry after marking with specific fluorescent antibodies (Luminex) and measured as a percentage.
Cycle 2, Group A : T4 DR+ lymphocytes BEFORE double filtration plasmapheresis | Day 0 Hour 0
  5 mL of blood will be collected in an EDTA tube BEFORE double filtration plasmapheresis and cell counts will be made by flow cytometry after marking with specific fluorescent antibodies (Luminex) and measured as a percentage.
Cycle 2, Group A : T8 lymphocytes BEFORE double filtration plasmapheresis | Day 0 Hour 0
  5 mL of blood will be collected in an EDTA tube BEFORE double filtration plasmapheresis and cell counts will be made by flow cytometry after marking with specific fluorescent antibodies (Luminex) and measured as a percentage.
Cycle 2, Group A : T8 DR+ lymphocytes BEFORE double filtration plasmapheresis | Day 0 Hour 0
  5 mL of blood will be collected in an EDTA tube BEFORE double filtration plasmapheresis and cell counts will be made by flow cytometry after marking with specific fluorescent antibodies (Luminex) and measured as a percentage.
Cycle 2, Group A : B lymphocytes BEFORE double filtration plasmapheresis | Day 0 Hour 0
  5 mL of blood will be collected in an EDTA tube BEFORE double filtration plasmapheresis and cell counts will be made by flow cytometry after marking with specific fluorescent antibodies (Luminex) a,d measured as a percentage.
Cycle 2, Group A : CD45RA+CCR7+ cells BEFORE double filtration plasmapheresis | Day 0 Hour 0
  5 mL of blood will be collected in an EDTA tube BEFORE double filtration plasmapheresis and cell counts will be made by flow cytometry after marking with specific fluorescent antibodies (Luminex) a,d measured as a percentage.
Cycle 2, Group A : CD45RA-CCR7+ cells BEFORE double filtration plasmapheresis | Day 0 Hour 0
  5 mL of blood will be collected in an EDTA tube BEFORE double filtration plasmapheresis and cell counts will be made by flow cytometry after marking with specific fluorescent antibodies (Luminex) a,d measured as a percentage.
Cycle 2, Group A : CD45RA-CCR7- cells BEFORE double filtration plasmapheresis | Day 0 Hour 0
  5 mL of blood will be collected in an EDTA tube BEFORE double filtration plasmapheresis and cell counts will be made by flow cytometry after marking with specific fluorescent antibodies (Luminex) a,d measured as a percentage.
Cycle 2, Group A : CCR6-CXCR3- cells BEFORE double filtration plasmapheresis | Day 0 Hour 0
  5 mL of blood will be collected in an EDTA tube BEFORE double filtration plasmapheresis and cell counts will be made by flow cytometry after marking with specific fluorescent antibodies (Luminex) a,d measured as a percentage.
Cycle 2, Group A : T4 lymphocytes AFTER double filtration plasmapheresis | Day 0 Hour 3
  5 mL of blood will be collected in an EDTA tube AFTER double filtration plasmapheresis and cell counts will be made by flow cytometry after marking with specific fluorescent antibodies (Luminex) a,d measured as a percentage.
Cycle 2, Group A : T4 DR+ lymphocytes AFTER double filtration plasmapheresis | Day 0 Hour 3
  5 mL of blood will be collected in an EDTA tube AFTER double filtration plasmapheresis and cell counts will be made by flow cytometry after marking with specific fluorescent antibodies (Luminex) and measured as a percentage.
Cycle 2, Group A : T8 lymphocytes AFTER double filtration plasmapheresis | Day 0 Hour 3
  5 mL of blood will be collected in an EDTA tube AFTER double filtration plasmapheresis and cell counts will be made by flow cytometry after marking with specific fluorescent antibodies (Luminex) and measured as a percentage.
Cycle 2, Group A : T8 DR+ lymphocytes AFTER double filtration plasmapheresis | Day 0 Hour 3
  5 mL of blood will be collected in an EDTA tube AFTER double filtration plasmapheresis and cell counts will be made by flow cytometry after marking with specific fluorescent antibodies (Luminex) and measured as a percentage.
Cycle 2, Group A : B lymphocytes AFTER double filtration plasmapheresis | Day 0 Hour 3
  5 mL of blood will be collected in an EDTA tube AFTER double filtration plasmapheresis and cell counts will be made by flow cytometry after marking with specific fluorescent antibodies (Luminex) and measured as a percentage.
Cycle 2, Group A : CD45RA+CCR7+ cells AFTER double filtration plasmapheresis | Day 0 Hour 3
  5 mL of blood will be collected in an EDTA tube AFTER double filtration plasmapheresis and cell counts will be made by flow cytometry after marking with specific fluorescent antibodies (Luminex) and measured as a percentage.
Cycle 2, Group A : CD45RA-CCR7+ cells AFTER double filtration plasmapheresis | Day 0 Hour 3
  5 mL of blood will be collected in an EDTA tube AFTER double filtration plasmapheresis and cell counts will be made by flow cytometry after marking with specific fluorescent antibodies (Luminex) and measured as a percentage.
Cycle 2, Group A : CD45RA-CCR7- cells AFTER double filtration plasmapheresis | Day 0 Hour 3
  5 mL of blood will be collected in an EDTA tube AFTER double filtration plasmapheresis and cell counts will be made by flow cytometry after marking with specific fluorescent antibodies (Luminex) and measured as a percentage.
Cycle 2, Group A : CCR6-CXCR3- cells AFTER double filtration plasmapheresis | Day 0 Hour 3
  5 mL of blood will be collected in an EDTA tube AFTER double filtration plasmapheresis and cell counts will be made by flow cytometry after marking with specific fluorescent antibodies (Luminex) and measured as a percentage.
Cycle 2, Group A : T4 lymphocytes 7-10 days AFTER double filtration plasmapheresis | Day 7 - 10
  5 mL of blood will be collected in an EDTA tube AFTER double filtration plasmapheresis and cell counts will be made by flow cytometry after marking with specific fluorescent antibodies (Luminex) and measured as a percentage.
Cycle 2, Group A : T4 DR+ lymphocytes 7-10 days AFTER double filtration plasmapheresis | Day 7 - 10
  5 mL of blood will be collected in an EDTA tube AFTER double filtration plasmapheresis and cell counts will be made by flow cytometry after marking with specific fluorescent antibodies (Luminex) and measured as a percentage.
Cycle 2, Group A : T8 lymphocytes 7-10 days AFTER double filtration plasmapheresis | Day 7 - 10
  5 mL of blood will be collected in an EDTA tube AFTER double filtration plasmapheresis and cell counts will be made by flow cytometry after marking with specific fluorescent antibodies (Luminex) and measured as a percentage.
Cycle 2, Group A : T8 DR+ lymphocytes 7-10 days AFTER double filtration plasmapheresis | Day 7 - 10
  5 mL of blood will be collected in an EDTA tube AFTER double filtration plasmapheresis and cell counts will be made by flow cytometry after marking with specific fluorescent antibodies (Luminex) and measured as a percentage.
Cycle 2, Group A : B lymphocytes 7-10 days AFTER double filtration plasmapheresis | Day 7 - 10
  5 mL of blood will be collected in an EDTA tube AFTER double filtration plasmapheresis and cell counts will be made by flow cytometry after marking with specific fluorescent antibodies (Luminex) and measured as a percentage.
Cycle 2, Group A : CD45RA+CCR7+ cells 7-10 days AFTER double filtration plasmapheresis | Day 7 - 10
  5 mL of blood will be collected in an EDTA tube AFTER double filtration plasmapheresis and cell counts will be made by flow cytometry after marking with specific fluorescent antibodies (Luminex) and measured as a percentage.
Cycle 2, Group A : CD45RA-CCR7+ cells 7-10 days AFTER double filtration plasmapheresis | Day 7 - 10
  5 mL of blood will be collected in an EDTA tube AFTER double filtration plasmapheresis and cell counts will be made by flow cytometry after marking with specific fluorescent antibodies (Luminex) and measured as a percentage.
Cycle 2, Group A : CD45RA-CCR7- cells 7-10 days AFTER double filtration plasmapheresis | Day 7 - 10
  5 mL of blood will be collected in an EDTA tube AFTER double filtration plasmapheresis and cell counts will be made by flow cytometry after marking with specific fluorescent antibodies (Luminex) and measured as a percentage.
Cycle 2, Group A : CCR6-CXCR3- cells 7-10 days AFTER double filtration plasmapheresis | Day 7 - 10
  5 mL of blood will be collected in an EDTA tube AFTER double filtration plasmapheresis and cell counts will be made by flow cytometry after marking with specific fluorescent antibodies (Luminex) and measured as a percentage.
Cycle 2, Group B : T4 lymphocytes BEFORE single plasma exchange | Day 0 Hour 0
  5 mL of blood will be collected in an EDTA tube BEFORE single plasma exchange and cell counts will be made by flow cytometry after marking with specific fluorescent antibodies (Luminex) and measured as a percentage.
Cycle 2, Group B : T4 DR+ lymphocytes BEFORE single plasma exchange | Day 0 Hour 0
  5 mL of blood will be collected in an EDTA tube BEFORE single plasma exchange and cell counts will be made by flow cytometry after marking with specific fluorescent antibodies (Luminex) and measured as a percentage.
Cycle 2, Group B : T8 lymphocytes BEFORE single plasma exchange | Day 0 Hour 0
  5 mL of blood will be collected in an EDTA tube BEFORE single plasma exchange and cell counts will be made by flow cytometry after marking with specific fluorescent antibodies (Luminex) and measured as a percentage.
Cycle 2, Group B : T8 DR+ lymphocytes BEFORE single plasma exchange | Day 0 Hour 0
  5 mL of blood will be collected in an EDTA tube BEFORE single plasma exchange and cell counts will be made by flow cytometry after marking with specific fluorescent antibodies (Luminex) and measured as a percentage.
Cycle 2, Group B : B lymphocytes BEFORE single plasma exchange | Day 0 Hour 0
  5 mL of blood will be collected in an EDTA tube BEFORE single plasma exchange and cell counts will be made by flow cytometry after marking with specific fluorescent antibodies (Luminex) and measured as a percentage.
Cycle 2, Group B : CD45RA+CCR7+ cells BEFORE single plasma exchange | Day 0 Hour 0
  5 mL of blood will be collected in an EDTA tube BEFORE single plasma exchange and cell counts will be made by flow cytometry after marking with specific fluorescent antibodies (Luminex) and measured as a percentage.
Cycle 2, Group B : CD45RA-CCR7+ cells BEFORE single plasma exchange | Day 0 Hour 0
  5 mL of blood will be collected in an EDTA tube BEFORE single plasma exchange and cell counts will be made by flow cytometry after marking with specific fluorescent antibodies (Luminex) and measured as a percentage.
Cycle 2, Group B : CD45RA-CCR7- cells BEFORE single plasma exchange | Day 0 Hour 0
  5 mL of blood will be collected in an EDTA tube BEFORE single plasma exchange and cell counts will be made by flow cytometry after marking with specific fluorescent antibodies (Luminex) and measured as a percentage.
Cycle 2, Group B : CCR6-CXCR3- cells BEFORE single plasma exchange | Day 0 Hour 0
  5 mL of blood will be collected in an EDTA tube BEFORE single plasma exchange and cell counts will be made by flow cytometry after marking with specific fluorescent antibodies (Luminex) and measured as a percentage.
Cycle 2, Group B : T4 lymphocytes AFTER single plasma exchange | Day 0 Hour 3
  5 mL of blood will be collected in an EDTA tube AFTER single plasma exchange and cell counts will be made by flow cytometry after marking with specific fluorescent antibodies (Luminex) and measured as a percentage.
Cycle 2, Group B : T4 DR+ lymphocytes AFTER single plasma exchange | Day 0 Hour 3
  5 mL of blood will be collected in an EDTA tube AFTER single plasma exchange and cell counts will be made by flow cytometry after marking with specific fluorescent antibodies (Luminex) and measured as a percentage.
Cycle 2, Group B : T8 lymphocytes AFTER single plasma exchange | Day 0 Hour 3
  5 mL of blood will be collected in an EDTA tube AFTER single plasma exchange and cell counts will be made by flow cytometry after marking with specific fluorescent antibodies (Luminex) and measured as a percentage.
Cycle 2, Group B : T8 DR+ lymphocytes AFTER single plasma exchange | Day 0 Hour 3
  5 mL of blood will be collected in an EDTA tube AFTER single plasma exchange and cell counts will be made by flow cytometry after marking with specific fluorescent antibodies (Luminex) and measured as a percentage.
Cycle 2, Group B : B lymphocytes AFTER single plasma exchange | Day 0 Hour 3
  5 mL of blood will be collected in an EDTA tube AFTER single plasma exchange and cell counts will be made by flow cytometry after marking with specific fluorescent antibodies (Luminex) and measured as a percentage.
Cycle 2, Group B : CD45RA+CCR7+ cells AFTER single plasma exchange | Day 0 Hour 3
  5 mL of blood will be collected in an EDTA tube AFTER single plasma exchange and cell counts will be made by flow cytometry after marking with specific fluorescent antibodies (Luminex) and measured as a percentage.
Cycle 2, Group B : CD45RA-CCR7+ cells AFTER single plasma exchange | Day 0 Hour 3
  5 mL of blood will be collected in an EDTA tube AFTER single plasma exchange and cell counts will be made by flow cytometry after marking with specific fluorescent antibodies (Luminex) and measured as a percentage.
Cycle 2, Group B : CD45RA-CCR7- cells AFTER single plasma exchange | Day 0 Hour 3
  5 mL of blood will be collected in an EDTA tube AFTER single plasma exchange and cell counts will be made by flow cytometry after marking with specific fluorescent antibodies (Luminex) and measured as a percentage.
Cycle 2, Group B : CCR6-CXCR3- cells AFTER single plasma exchange | Day 0 Hour 3
  5 mL of blood will be collected in an EDTA tube AFTER single plasma exchange and cell counts will be made by flow cytometry after marking with specific fluorescent antibodies (Luminex) and measured as a percentage.
Cycle 2, Group B : T4 lymphocytes 7-10 days AFTER single plasma exchange | Day 7-10
  5 mL of blood will be collected in an EDTA tube AFTER single plasma exchange and cell counts will be made by flow cytometry after marking with specific fluorescent antibodies (Luminex) and measured as a percentage.
Cycle 2, Group B : T4 DR+ lymphocytes 7-10 days AFTER single plasma exchange | Day 7-10
  5 mL of blood will be collected in an EDTA tube AFTER single plasma exchange and cell counts will be made by flow cytometry after marking with specific fluorescent antibodies (Luminex) and measured as a percentage.
Cycle 2, Group B : T8 lymphocytes 7-10 days AFTER single plasma exchange | Day 7-10
  5 mL of blood will be collected in an EDTA tube AFTER single plasma exchange and cell counts will be made by flow cytometry after marking with specific fluorescent antibodies (Luminex) and measured as a percentage.
Cycle 2, Group B : T8 DR+ lymphocytes 7-10 days AFTER single plasma exchange | Day 7-10
  5 mL of blood will be collected in an EDTA tube AFTER single plasma exchange and cell counts will be made by flow cytometry after marking with specific fluorescent antibodies (Luminex) and measured as a percentage.
Cycle 2, Group B : B lymphocytes 7-10 days AFTER single plasma exchange | Day 7-10
  5 mL of blood will be collected in an EDTA tube AFTER single plasma exchange and cell counts will be made by flow cytometry after marking with specific fluorescent antibodies (Luminex) and measured as a percentage.
Cycle 2, Group B : CD45RA+CCR7+ cells 7-10 days AFTER single plasma exchange | Day 7-10
  5 mL of blood will be collected in an EDTA tube AFTER single plasma exchange and cell counts will be made by flow cytometry after marking with specific fluorescent antibodies (Luminex) and measured as a percentage.
Cycle 2, Group B : CD45RA-CCR7+ cells 7-10 days AFTER single plasma exchange | Day 7-10
  5 mL of blood will be collected in an EDTA tube AFTER single plasma exchange and cell counts will be made by flow cytometry after marking with specific fluorescent antibodies (Luminex) and measured as a percentage.
Cycle 2, Group B : CD45RA-CCR7- cells 7-10 days AFTER single plasma exchange | Day 7-10
  5 mL of blood will be collected in an EDTA tube AFTER single plasma exchange and cell counts will be made by flow cytometry after marking with specific fluorescent antibodies (Luminex) and measured a percentage.
Cycle 2, Group B : CCR6-CXCR3- cells 7-10 days AFTER single plasma exchange | Day 7-10
  5 mL of blood will be collected in an EDTA tube AFTER single plasma exchange and cell counts will be made by flow cytometry after marking with specific fluorescent antibodies (Luminex) and measured as a percentage.
Cycle 3, Group A : T4 lymphocytes BEFORE single plasma exchange | Day 0 Hour 0
  5 mL of blood will be collected in an EDTA tube BEFORE single plasma exchange and cell counts will be made by flow cytometry after marking with specific fluorescent antibodies (Luminex) and measured as a percentage.
Cycle 3, Group A : T4 DR+ lymphocytes BEFORE single plasma exchange | Day 0 Hour 0
  5 mL of blood will be collected in an EDTA tube BEFORE single plasma exchange and cell counts will be made by flow cytometry after marking with specific fluorescent antibodies (Luminex) and measured as a percentage.
Cycle 3, Group A : T8 lymphocytes BEFORE single plasma exchange | Day 0 Hour 0
  5 mL of blood will be collected in an EDTA tube BEFORE single plasma exchange and cell counts will be made by flow cytometry after marking with specific fluorescent antibodies (Luminex) and measured as a percentage.
Cycle 3, Group A : T8 DR+ lymphocytes BEFORE single plasma exchange | Day 0 Hour 0
  5 mL of blood will be collected in an EDTA tube BEFORE single plasma exchange and cell counts will be made by flow cytometry after marking with specific fluorescent antibodies (Luminex) and measured as a percentage.
Cycle 3, Group A : B lymphocytes BEFORE single plasma exchange | Day 0 Hour 0
  5 mL of blood will be collected in an EDTA tube BEFORE single plasma exchange and cell counts will be made by flow cytometry after marking with specific fluorescent antibodies (Luminex) and measured as a percentage.
Cycle 3, Group A : CC45RA+CCR7+ cells BEFORE single plasma exchange | Day 0 Hour 0
  5 mL of blood will be collected in an EDTA tube BEFORE single plasma exchange and cell counts will be made by flow cytometry after marking with specific fluorescent antibodies (Luminex) and measured as a percentage.
Cycle 3, Group A : CC45RA-CCR7+ cells BEFORE single plasma exchange | Day 0 Hour 0
  5 mL of blood will be collected in an EDTA tube BEFORE single plasma exchange and cell counts will be made by flow cytometry after marking with specific fluorescent antibodies (Luminex) and measured as a percentage.
Cycle 3, Group A : CC45RA-CCR7- cells BEFORE single plasma exchange | Day 0 Hour 0
  5 mL of blood will be collected in an EDTA tube BEFORE single plasma exchange and cell counts will be made by flow cytometry after marking with specific fluorescent antibodies (Luminex) and measured as a percentage.
Cycle 3, Group A : CCR6-CXCR3- cells BEFORE single plasma exchange | Day 0 Hour 0
  5 mL of blood will be collected in an EDTA tube BEFORE single plasma exchange and cell counts will be made by flow cytometry after marking with specific fluorescent antibodies (Luminex) and measured as a percentage.
Cycle 3, Group A : T4 lymphocytes AFTER single plasma exchange | Day 0 Hour 3
  5 mL of blood will be collected in an EDTA tube AFTER single plasma exchange and cell counts will be made by flow cytometry after marking with specific fluorescent antibodies (Luminex) and measured as a percentage.
Cycle 3, Group A : T4 DR+ lymphocytes AFTER single plasma exchange | Day 0 Hour 3
  5 mL of blood will be collected in an EDTA tube AFTER single plasma exchange and cell counts will be made by flow cytometry after marking with specific fluorescent antibodies (Luminex) and measured as a percentage.
Cycle 3, Group A : T8 lymphocytes AFTER single plasma exchange | Day 0 Hour 3
  5 mL of blood will be collected in an EDTA tube AFTER single plasma exchange and cell counts will be made by flow cytometry after marking with specific fluorescent antibodies (Luminex) and measured as a percentage.
Cycle 3, Group A : T8 DR+ lymphocytes AFTER single plasma exchange | Day 0 Hour 3
  5 mL of blood will be collected in an EDTA tube AFTER single plasma exchange and cell counts will be made by flow cytometry after marking with specific fluorescent antibodies (Luminex) and measured as a percentage.
Cycle 3, Group A : B lymphocytes AFTER single plasma exchange | Day 0 Hour 3
  5 mL of blood will be collected in an EDTA tube AFTER single plasma exchange and cell counts will be made by flow cytometry after marking with specific fluorescent antibodies (Luminex) and measured as a percentage.
Cycle 3, Group A : CD45RA+CCR7+ cells AFTER single plasma exchange | Day 0 Hour 3
  5 mL of blood will be collected in an EDTA tube AFTER single plasma exchange and cell counts will be made by flow cytometry after marking with specific fluorescent antibodies (Luminex) and measured as a percentage.
Cycle 3, Group A : CD45RA-CCR7+ cells AFTER single plasma exchange | Day 0 Hour 3
  5 mL of blood will be collected in an EDTA tube AFTER single plasma exchange and cell counts will be made by flow cytometry after marking with specific fluorescent antibodies (Luminex) and measured as a percentage.
Cycle 3, Group A : CD45RA-CCR7- cells AFTER single plasma exchange | Day 0 Hour 3
  5 mL of blood will be collected in an EDTA tube AFTER single plasma exchange and cell counts will be made by flow cytometry after marking with specific fluorescent antibodies (Luminex) and measured as a percentage.
Cycle 3, Group A : CCR6-CXCR3- cells AFTER single plasma exchange | Day 0 Hour 3
  5 mL of blood will be collected in an EDTA tube AFTER single plasma exchange and cell counts will be made by flow cytometry after marking with specific fluorescent antibodies (Luminex) and measured as a percentage.
Cycle 3, Group A : T4 DR+ lymphocytes 7-10 days AFTER single plasma exchange | Day 7-10
  5 mL of blood will be collected in an EDTA tube AFTER single plasma exchange and cell counts will be made by flow cytometry after marking with specific fluorescent antibodies (Luminex) and measured as a percentage.
Cycle 3, Group A : T4 lymphocytes 7 -10 days AFTER single plasma exchange | Day 7-10
  5 mL of blood will be collected in an EDTA tube AFTER single plasma exchange and cell counts will be made by flow cytometry after marking with specific fluorescent antibodies (Luminex) and measured as a percentage.
Cycle 3, Group A : T8 lymphocytes 7-10 days AFTER single plasma exchange | Day 7-10
  5 mL of blood will be collected in an EDTA tube AFTER single plasma exchange and cell counts will be made by flow cytometry after marking with specific fluorescent antibodies (Luminex) and measured as a percentage.
Cycle 3, Group A : T8 DR+ lymphocytes 7-10 days AFTER single plasma exchange | Day 7-10
  5 mL of blood will be collected in an EDTA tube AFTER single plasma exchange and cell counts will be made by flow cytometry after marking with specific fluorescent antibodies (Luminex) and measured as a percentage.
Cycle 3, Group A : B lymphocytes 7-10 days AFTER single plasma exchange | Day 7-10
  5 mL of blood will be collected in an EDTA tube AFTER single plasma exchange and cell counts will be made by flow cytometry after marking with specific fluorescent antibodies (Luminex) and measured as a percentage.
Cycle 3, Group A : CD45RA+CCR7+ cells 7-10 days AFTER single plasma exchange | Day 7-10
  5 mL of blood will be collected in an EDTA tube AFTER single plasma exchange and cell counts will be made by flow cytometry after marking with specific fluorescent antibodies (Luminex) and measured as a percentage.
Cycle 3, Group A : CD45RA-CCR7+ cells 7-10 days AFTER single plasma exchange | Day 7-10
  5 mL of blood will be collected in an EDTA tube AFTER single plasma exchange and cell counts will be made by flow cytometry after marking with specific fluorescent antibodies (Luminex) and measured as a percentage.
Cycle 3, Group A : CD45RA-CCR7- cells 7-10 days AFTER single plasma exchange | Day 7-10
  5 mL of blood will be collected in an EDTA tube AFTER single plasma exchange and cell counts will be made by flow cytometry after marking with specific fluorescent antibodies (Luminex) and measured as a percentage.
Cycle 3, Group A : CCR6-CXCR3- cells 7-10 days AFTER single plasma exchange | Day 7-10
  5 mL of blood will be collected in an EDTA tube AFTER single plasma exchange and cell counts will be made by flow cytometry after marking with specific fluorescent antibodies (Luminex) and measured as a percentage.
Cycle 3, Group B : T4 lymphocytes BEFORE double filtration plasmapheresis | Day 0 Hour 0
  5 mL of blood will be collected in an EDTA tube BEFORE double filtration and cell counts will be made by flow cytometry after marking with specific fluorescent antibodies (Luminex) and measured as a percentage.
Cycle 3, Group B : T4 DR+ lymphocytes BEFORE double filtration plasmapheresis | Day 0 Hour 0
  5 mL of blood will be collected in an EDTA tube BEFORE double filtration and cell counts will be made by flow cytometry after marking with specific fluorescent antibodies (Luminex) and measured as a percentage.
Cycle 3, Group B : T8 lymphocytes BEFORE double filtration plasmapheresis | Day 0 Hour 0
  5 mL of blood will be collected in an EDTA tube BEFORE double filtration and cell counts will be made by flow cytometry after marking with specific fluorescent antibodies (Luminex) and measured as a percentage.
Cycle 3, Group B : T8 DR+ lymphocytes BEFORE double filtration plasmapheresis | Day 0 Hour 0
  5 mL of blood will be collected in an EDTA tube BEFORE double filtration and cell counts will be made by flow cytometry after marking with specific fluorescent antibodies (Luminex) and measured as a percentage.
Cycle 3, Group B : B lymphocytes BEFORE double filtration plasmapheresis | Day 0 Hour 0
  5 mL of blood will be collected in an EDTA tube BEFORE double filtration and cell counts will be made by flow cytometry after marking with specific fluorescent antibodies (Luminex) and measured as a percentage.
Cycle 3, Group B : CD45RA+CCR7+ cells BEFORE double filtration plasmapheresis | Day 0 Hour 0
  5 mL of blood will be collected in an EDTA tube BEFORE double filtration and cell counts will be made by flow cytometry after marking with specific fluorescent antibodies (Luminex) and measured as a percentage.
Cycle 3, Group B : CD45RA-CCR7+ cells BEFORE double filtration plasmapheresis | Day 0 Hour 0
  5 mL of blood will be collected in an EDTA tube BEFORE double filtration and cell counts will be made by flow cytometry after marking with specific fluorescent antibodies (Luminex) and measured as a percentage.
Cycle 3, Group B : CD45RA-CCR7- cells BEFORE double filtration plasmapheresis | Day 0 Hour 0
  5 mL of blood will be collected in an EDTA tube BEFORE double filtration and cell counts will be made by flow cytometry after marking with specific fluorescent antibodies (Luminex) and measured as a percentage.
Cycle 3, Group B : CCR6-CXCR3- cells BEFORE double filtration plasmapheresis | Day 0 Hour 0
  5 mL of blood will be collected in an EDTA tube BEFORE double filtration and cell counts will be made by flow cytometry after marking with specific fluorescent antibodies (Luminex) and measured as a percentage.
Cycle 3, Group B : T4 lymphocytes AFTER double filtration plasmapheresis | Day 0 Hour 3
  5 mL of blood will be collected in an EDTA tube AFTER double filtration and cell counts will be made by flow cytometry after marking with specific fluorescent antibodies (Luminex) and measured as a percentage.
Cycle 3, Group B : T4 DR+ lymphocytes AFTER double filtration plasmapheresis | Day 0 Hour 3
  5 mL of blood will be collected in an EDTA tube AFTER double filtration and cell counts will be made by flow cytometry after marking with specific fluorescent antibodies (Luminex) and measured as a percentage.
Cycle 3, Group B : T8 lymphocytes AFTER double filtration plasmapheresis | Day 0 Hour 3
  5 mL of blood will be collected in an EDTA tube AFTER double filtration and cell counts will be made by flow cytometry after marking with specific fluorescent antibodies (Luminex) and measured as a percentage.
Cycle 3, Group B : T8 DR+ lymphocytes AFTER double filtration plasmapheresis | Day 0 Hour 3
  5 mL of blood will be collected in an EDTA tube AFTER double filtration and cell counts will be made by flow cytometry after marking with specific fluorescent antibodies (Luminex) and measured as a percentage.
Cycle 3, Group B : B lymphocytes AFTER double filtration plasmapheresis | Day 0 Hour 3
  5 mL of blood will be collected in an EDTA tube AFTER double filtration and cell counts will be made by flow cytometry after marking with specific fluorescent antibodies (Luminex) and measured as a percentage.
Cycle 3, Group B : CD45RA+CCR7+ cells AFTER double filtration plasmapheresis | Day 0 Hour 3
  5 mL of blood will be collected in an EDTA tube AFTER double filtration and cell counts will be made by flow cytometry after marking with specific fluorescent antibodies (Luminex) and measured as a percentage.
Cycle 3, Group B : CD45RA-CCR7+ cells AFTER double filtration plasmapheresis | Day 0 Hour 3
  5 mL of blood will be collected in an EDTA tube AFTER double filtration and cell counts will be made by flow cytometry after marking with specific fluorescent antibodies (Luminex) and measured as a percentage.
Cycle 3, Group B : CD45RA-CCR7- cells AFTER double filtration plasmapheresis | Day 0 Hour 3
  5 mL of blood will be collected in an EDTA tube AFTER double filtration and cell counts will be made by flow cytometry after marking with specific fluorescent antibodies (Luminex) and measured as a percentage.
Cycle 3, Group B : CCR6-CXCR3- cells AFTER double filtration plasmapheresis | Day 0 Hour 3
  5 mL of blood will be collected in an EDTA tube AFTER double filtration and cell counts will be made by flow cytometry after marking with specific fluorescent antibodies (Luminex) and measured as a percentage.
Cycle 3, Group B : T4 lymphocytes 7-10 days AFTER double filtration plasmapheresis | Day 7-10
  5 mL of blood will be collected in an EDTA tube AFTER double filtration and cell counts will be made by flow cytometry after marking with specific fluorescent antibodies (Luminex) and measured as a percentage.
Cycle 3, Group B : T4 DR+ lymphocytes 7-10 days AFTER double filtration plasmapheresis | Day 7-10
  5 mL of blood will be collected in an EDTA tube AFTER double filtration and cell counts will be made by flow cytometry after marking with specific fluorescent antibodies (Luminex) and measured as a percentage.
Cycle 3, Group B : T8 lymphocytes 7-10 days AFTER double filtration plasmapheresis | Day 7-10
  5 mL of blood will be collected in an EDTA tube AFTER double filtration and cell counts will be made by flow cytometry after marking with specific fluorescent antibodies (Luminex) and measured as a percentage.
Cycle 3, Group B : T8 DR+ lymphocytes 7-10 days AFTER double filtration plasmapheresis | Day 7-10
  5 mL of blood will be collected in an EDTA tube AFTER double filtration and cell counts will be made by flow cytometry after marking with specific fluorescent antibodies (Luminex) and measured as a percentage.
Cycle 3, Group B : B lymphocytes 7-10 days AFTER double filtration plasmapheresis | Day 7-10
  5 mL of blood will be collected in an EDTA tube AFTER double filtration and cell counts will be made by flow cytometry after marking with specific fluorescent antibodies (Luminex) and measured as a percentage.
Cycle 3, Group B : CD45RA+CCR7+ cells 7-10 days AFTER double filtration plasmapheresis | Day 7-10
  5 mL of blood will be collected in an EDTA tube AFTER double filtration and cell counts will be made by flow cytometry after marking with specific fluorescent antibodies (Luminex) and measured as a percentage.
Cycle 3, Group B : CD45RA-CCR7+ cells 7-10 days AFTER double filtration plasmapheresis | Day 7-10
  5 mL of blood will be collected in an EDTA tube AFTER double filtration and cell counts will be made by flow cytometry after marking with specific fluorescent antibodies (Luminex) and measured as a percentage.
Cycle 3, Group B : CD45RA-CCR7- cells 7-10 days AFTER double filtration plasmapheresis | Day 7-10
  5 mL of blood will be collected in an EDTA tube AFTER double filtration and cell counts will be made by flow cytometry after marking with specific fluorescent antibodies (Luminex) and measured as a percentage.
Cycle 3, Group B : CCR6-CXCR3- cells 7-10 days AFTER double filtration plasmapheresis | Day 7-10
  5 mL of blood will be collected in an EDTA tube AFTER double filtration and cell counts will be made by flow cytometry after marking with specific fluorescent antibodies (Luminex) and measured as a percentage.
Cycle 4, Group A : T4 lymphocytes BEFORE double filtration plasmapheresis | Day 0 Hour 0
  5 mL of blood will be collected in an EDTA tube BEFORE double filtration and cell counts will be made by flow cytometry after marking with specific fluorescent antibodies (Luminex) and measured as a percentage.
Cycle 4, Group A : T4 DR+ lymphocytes BEFORE double filtration plasmapheresis | Day 0 Hour 0
  5 mL of blood will be collected in an EDTA tube BEFORE double filtration and cell counts will be made by flow cytometry after marking with specific fluorescent antibodies (Luminex) and measured as a percentage.
Cycle 4, Group A : T8 lymphocytes BEFORE double filtration plasmapheresis | Day 0 Hour 0
  5 mL of blood will be collected in an EDTA tube BEFORE double filtration and cell counts will be made by flow cytometry after marking with specific fluorescent antibodies (Luminex) and measured as a percentage.
Cycle 4, Group A : T8 DR+ lymphocytes BEFORE double filtration plasmapheresis | Day 0 Hour 0
  5 mL of blood will be collected in an EDTA tube BEFORE double filtration and cell counts will be made by flow cytometry after marking with specific fluorescent antibodies (Luminex) and measured as a percentage.
Cycle 4, Group A : B lymphocytes BEFORE double filtration plasmapheresis | Day 0 Hour 0
  5 mL of blood will be collected in an EDTA tube BEFORE double filtration and cell counts will be made by flow cytometry after marking with specific fluorescent antibodies (Luminex) and measured as a percentage.
Cycle 4, Group A : CD45RA+CCR7+ cells BEFORE double filtration plasmapheresis | Day 0 Hour 0
  5 mL of blood will be collected in an EDTA tube BEFORE double filtration and cell counts will be made by flow cytometry after marking with specific fluorescent antibodies (Luminex) and measured as a percentage.
Cycle 4, Group A : CD45RA-CCR7+ cells BEFORE double filtration plasmapheresis | Day 0 Hour 0
  5 mL of blood will be collected in an EDTA tube BEFORE double filtration and cell counts will be made by flow cytometry after marking with specific fluorescent antibodies (Luminex) and measured as a percentage.
Cycle 4, Group A : CD45RA-CCR7- cells BEFORE double filtration plasmapheresis | Day 0 Hour 0
  5 mL of blood will be collected in an EDTA tube BEFORE double filtration and cell counts will be made by flow cytometry after marking with specific fluorescent antibodies (Luminex) and measured as a percentage.
Cycle 4, Group A : CCR6-CXCR3- cells BEFORE double filtration plasmapheresis | Day 0 Hour 0
  5 mL of blood will be collected in an EDTA tube BEFORE double filtration and cell counts will be made by flow cytometry after marking with specific fluorescent antibodies (Luminex) and measured as a percentage.
Cycle 4, Group A : T4 lymphocytes AFTER double filtration plasmapheresis | Day 0 Hour 3
  5 mL of blood will be collected in an EDTA tube AFTER double filtration and cell counts will be made by flow cytometry after marking with specific fluorescent antibodies (Luminex) and measured as a percentage.
Cycle 4, Group A : T4 DR+ lymphocytes AFTER double filtration plasmapheresis | Day 0 Hour 3
  5 mL of blood will be collected in an EDTA tube AFTER double filtration and cell counts will be made by flow cytometry after marking with specific fluorescent antibodies (Luminex) and measured as a percentage.
Cycle 4, Group A : T8 lymphocytes AFTER double filtration plasmapheresis | Day 0 Hour 3
  5 mL of blood will be collected in an EDTA tube AFTER double filtration and cell counts will be made by flow cytometry after marking with specific fluorescent antibodies (Luminex) and measured as a percentage.
Cycle 4, Group A : T8 DR+ lymphocytes AFTER double filtration plasmapheresis | Day 0 Hour 3
  5 mL of blood will be collected in an EDTA tube AFTER double filtration and cell counts will be made by flow cytometry after marking with specific fluorescent antibodies (Luminex) and measured as a percentage.
Cycle 4, Group A : B lymphocytes AFTER double filtration plasmapheresis | Day 0 Hour 3
  5 mL of blood will be collected in an EDTA tube AFTER double filtration and cell counts will be made by flow cytometry after marking with specific fluorescent antibodies (Luminex) and measured as a percentage.
Cycle 4, Group A : CD45RA+CCR7+ cells AFTER double filtration plasmapheresis | Day 0 Hour 3
  5 mL of blood will be collected in an EDTA tube AFTER double filtration and cell counts will be made by flow cytometry after marking with specific fluorescent antibodies (Luminex) and measured as a percentage.
Cycle 4, Group A : CD45RA-CCR7+ cells AFTER double filtration plasmapheresis | Day 0 Hour 3
  5 mL of blood will be collected in an EDTA tube AFTER double filtration and cell counts will be made by flow cytometry after marking with specific fluorescent antibodies (Luminex) and measured as a percentage.
Cycle 4, Group A : CD45RA-CCR7- cells AFTER double filtration plasmapheresis | Day 0 Hour 3
  5 mL of blood will be collected in an EDTA tube AFTER double filtration and cell counts will be made by flow cytometry after marking with specific fluorescent antibodies (Luminex) and measured as a percentage.
Cycle 4, Group A : CCR6-CXCR3- cells AFTER double filtration plasmapheresis | Day 0 Hour 3
  5 mL of blood will be collected in an EDTA tube AFTER double filtration and cell counts will be made by flow cytometry after marking with specific fluorescent antibodies (Luminex) and measured as a percentage.
Cycle 4, Group A : T4 lymphocytes 7-10 days AFTER double filtration plasmapheresis | Day 7-10
  5 mL of blood will be collected in an EDTA tube AFTER double filtration and cell counts will be made by flow cytometry after marking with specific fluorescent antibodies (Luminex) and measured as a percentage.
Cycle 4, Group A : T4 DR+ lymphocytes 7-10 days AFTER double filtration plasmapheresis | Day 7-10
  5 mL of blood will be collected in an EDTA tube AFTER double filtration and cell counts will be made by flow cytometry after marking with specific fluorescent antibodies (Luminex) and measured as a percentage.
Cycle 4, Group A : T8 lymphocytes 7-10 days AFTER double filtration plasmapheresis | Day 7-10
  5 mL of blood will be collected in an EDTA tube AFTER double filtration and cell counts will be made by flow cytometry after marking with specific fluorescent antibodies (Luminex) and measured as a percentage.
Cycle 4, Group A : T8 DR+ lymphocytes 7-10 days AFTER double filtration plasmapheresis | Day 7-10
  5 mL of blood will be collected in an EDTA tube AFTER double filtration and cell counts will be made by flow cytometry after marking with specific fluorescent antibodies (Luminex) and measured as a percentage.
Cycle 4, Group A : B lymphocytes 7-10 days AFTER double filtration plasmapheresis | Day 7-10
  5 mL of blood will be collected in an EDTA tube AFTER double filtration and cell counts will be made by flow cytometry after marking with specific fluorescent antibodies (Luminex) and measured as a percentage.
Cycle 4, Group A : CD45RA+CCR7+ cells 7-10 days AFTER double filtration plasmapheresis | Day 7-10
  5 mL of blood will be collected in an EDTA tube AFTER double filtration and cell counts will be made by flow cytometry after marking with specific fluorescent antibodies (Luminex) and measured as a percentage.
Cycle 4, Group A : CD45RA-CCR7+ cells 7-10 days AFTER double filtration plasmapheresis | Day 7-10
  5 mL of blood will be collected in an EDTA tube AFTER double filtration and cell counts will be made by flow cytometry after marking with specific fluorescent antibodies (Luminex) and measured as a percentage.
Cycle 4, Group A : CD45RA-CCR7- cells 7-10 days AFTER double filtration plasmapheresis | Day 7-10
  5 mL of blood will be collected in an EDTA tube AFTER double filtration and cell counts will be made by flow cytometry after marking with specific fluorescent antibodies (Luminex) and measured as a percentage.
Cycle 4, Group A : CCR6-CXCR3- cells 7-10 days AFTER double filtration plasmapheresis | Day 7-10
  5 mL of blood will be collected in an EDTA tube AFTER double filtration and cell counts will be made by flow cytometry after marking with specific fluorescent antibodies (Luminex) and measured as a percentage.
Cycle 4, Group B : T4 lymphocytes BEFORE plasma exchange | Day 0 Hour 0
  5 mL of blood will be collected in an EDTA tube BEFORE single plasma exchange and cell counts will be made by flow cytometry after marking with specific fluorescent antibodies (Luminex) and measured as a percentage.
Cycle 4, Group B : T4 DR+ lymphocytes BEFORE plasma exchange | Day 0 Hour 0
  5 mL of blood will be collected in an EDTA tube BEFORE single plasma exchange and cell counts will be made by flow cytometry after marking with specific fluorescent antibodies (Luminex) and measured as a percentage.
Cycle 4, Group B : T8 lymphocytes BEFORE plasma exchange | Day 0 Hour 0
  5 mL of blood will be collected in an EDTA tube BEFORE single plasma exchange and cell counts will be made by flow cytometry after marking with specific fluorescent antibodies (Luminex) and measured as a percentage.
Cycle 4, Group B : T8 DR+ lymphocytes BEFORE single plasma exchange | Day 0 Hour 0
  5 mL of blood will be collected in an EDTA tube BEFORE single plasma exchange and cell counts will be made by flow cytometry after marking with specific fluorescent antibodies (Luminex) and measured as a percentage.
Cycle 4, Group B : B lymphocytes BEFORE single plasma exchange | Day 0 Hour 0
  5 mL of blood will be collected in an EDTA tube BEFORE single plasma exchange and cell counts will be made by flow cytometry after marking with specific fluorescent antibodies (Luminex) and measured as a percentage.
Cycle 4, Group B : CD45RA+CCR7+ cells BEFORE single plasma exchange | Day 0 Hour 0
  5 mL of blood will be collected in an EDTA tube BEFORE single plasma exchange and cell counts will be made by flow cytometry after marking with specific fluorescent antibodies (Luminex) and measured as a percentage.
Cycle 4, Group B : CD45RA-CCR7+ cells BEFORE single plasma exchange | Day 0 Hour 0
  5 mL of blood will be collected in an EDTA tube BEFORE single plasma exchange and cell counts will be made by flow cytometry after marking with specific fluorescent antibodies (Luminex) and measured as a percentage.
Cycle 4, Group B : CD45RA-CCR7- cells BEFORE single plasma exchange | Day 0 Hour 0
  5 mL of blood will be collected in an EDTA tube BEFORE single plasma exchange and cell counts will be made by flow cytometry after marking with specific fluorescent antibodies (Luminex) and measured as a percentage.
Cycle 4, Group B : CCR6-CXCR3- cells BEFORE single plasma exchange | Day 0 Hour 0
  5 mL of blood will be collected in an EDTA tube BEFORE single plasma exchange and cell counts will be made by flow cytometry after marking with specific fluorescent antibodies (Luminex) and measured as a percentage.
Cycle 4, Group B : T4 lymphocytes AFTER single plasma exchange | Day 0 Hour 3
  5 mL of blood will be collected in an EDTA tube AFTER single plasma exchange and cell counts will be made by flow cytometry after marking with specific fluorescent antibodies (Luminex) and measured as a percentage.
Cycle 4, Group B : T4 DR+ lymphocytes AFTER single plasma exchange | Day 0 Hour 3
  5 mL of blood will be collected in an EDTA tube AFTER single plasma exchange and cell counts will be made by flow cytometry after marking with specific fluorescent antibodies (Luminex) and measured as a percentage.
Cycle 4, Group B : T8 lymphocytes AFTER single plasma exchange | Day 0 Hour 3
  5 mL of blood will be collected in an EDTA tube AFTER single plasma exchange and cell counts will be made by flow cytometry after marking with specific fluorescent antibodies (Luminex) and measured as a percentage.
Cycle 4, Group B : T8 DR+ lymphocytes AFTER single plasma exchange | Day 0 Hour 3
  5 mL of blood will be collected in an EDTA tube AFTER single plasma exchange and cell counts will be made by flow cytometry after marking with specific fluorescent antibodies (Luminex) and measured as a percentage.
Cycle 4, Group B : B lymphocytes AFTER single plasma exchange | Day 0 Hour 3
  5 mL of blood will be collected in an EDTA tube AFTER single plasma exchange and cell counts will be made by flow cytometry after marking with specific fluorescent antibodies (Luminex) and measured as a percentage.
Cycle 4, Group B : CD45RA+CCR7+ cells AFTER single plasma exchange | Day 0 Hour 3
  5 mL of blood will be collected in an EDTA tube AFTER single plasma exchange and cell counts will be made by flow cytometry after marking with specific fluorescent antibodies (Luminex) and measured as a percentage.
Cycle 4, Group B : CD45RA-CCR7+ cells AFTER single plasma exchange | Day 0 Hour 3
  5 mL of blood will be collected in an EDTA tube AFTER single plasma exchange and cell counts will be made by flow cytometry after marking with specific fluorescent antibodies (Luminex) and measured as a percentage.
Cycle 4, Group B : CD45RA-CCR7- cells AFTER single plasma exchange | Day 0 Hour 3
  5 mL of blood will be collected in an EDTA tube AFTER single plasma exchange and cell counts will be made by flow cytometry after marking with specific fluorescent antibodies (Luminex) and measured as a percentage.
Cycle 4, Group B : CCR6-CXCR3- cells AFTER single plasma exchange | Day 0 Hour 3
  5 mL of blood will be collected in an EDTA tube AFTER single plasma exchange and cell counts will be made by flow cytometry after marking with specific fluorescent antibodies (Luminex) and measured as a percentage.
Cycle 4, Group B : T4 lymphocytes 7-10 days AFTER single plasma exchange | Day 7-10
  5 mL of blood will be collected in an EDTA tube AFTER single plasma exchange and cell counts will be made by flow cytometry after marking with specific fluorescent antibodies (Luminex) and measured as a percentage.
Cycle 4, Group B : T4 DR+ lymphocytes 7-10 days AFTER single plasma exchange | Day 7-10
  5 mL of blood will be collected in an EDTA tube AFTER single plasma exchange and cell counts will be made by flow cytometry after marking with specific fluorescent antibodies (Luminex) and measured as a percentage.
Cycle 4, Group B : T8 lymphocytes 7-10 days AFTER single plasma exchange | Day 7-10
  5 mL of blood will be collected in an EDTA tube AFTER single plasma exchange and cell counts will be made by flow cytometry after marking with specific fluorescent antibodies (Luminex) and measured as a percentage.
Cycle 4, Group B : T8 DR+ lymphocytes 7-10 days AFTER single plasma exchange | Day 7-10
  5 mL of blood will be collected in an EDTA tube AFTER single plasma exchange and cell counts will be made by flow cytometry after marking with specific fluorescent antibodies (Luminex) and measured as a percentage.
Cycle 4, Group B : B lymphocytes 7-10 days AFTER single plasma exchange | Day 7-10
  5 mL of blood will be collected in an EDTA tube AFTER single plasma exchange and cell counts will be made by flow cytometry after marking with specific fluorescent antibodies (Luminex) and measured as a percentage.
Cycle 4, Group B : CD45RA+CCR7+ cells 7-10 days AFTER single plasma exchange | Day 7-10
  5 mL of blood will be collected in an EDTA tube AFTER single plasma exchange and cell counts will be made by flow cytometry after marking with specific fluorescent antibodies (Luminex) and measured as a percentage.
Cycle 4, Group B : CD45RA-CCR7+ cells 7-10 days AFTER single plasma exchange | Day 7-10
  5 mL of blood will be collected in an EDTA tube AFTER single plasma exchange and cell counts will be made by flow cytometry after marking with specific fluorescent antibodies (Luminex) and measured as a percentage.
Cycle 4, Group B : CD45RA-CCR7- cells 7-10 days AFTER single plasma exchange | Day 7-10
  5 mL of blood will be collected in an EDTA tube AFTER single plasma exchange and cell counts will be made by flow cytometry after marking with specific fluorescent antibodies (Luminex) and measured as a percentage.
Cycle 4, Group B : CCR6-CXCR3- cells 7-10 days AFTER single plasma exchange | Day 7-10
  5 mL of blood will be collected in an EDTA tube AFTER single plasma exchange and cell counts will be made by flow cytometry after marking with specific fluorescent antibodies (Luminex) and measured as a percentage.
Cycle 5, Group A : T4 lymphocytes BEFORE single plasma exchange | Day 0, Hour 0
  5 mL of blood will be collected in an EDTA tube BEFORE single plasma exchange and cell counts will be made by flow cytometry after marking with specific fluorescent antibodies (Luminex) and measured as a percentage.
Cycle 5, Group A : T4 DR+ lymphocytes BEFORE single plasma exchange | Day 0, Hour 0
  5 mL of blood will be collected in an EDTA tube BEFORE single plasma exchange and cell counts will be made by flow cytometry after marking with specific fluorescent antibodies (Luminex) and measured as a percentage.
Cycle 5, Group A : T8 lymphocytes BEFORE single plasma exchange | Day 0, Hour 0
  5 mL of blood will be collected in an EDTA tube BEFORE single plasma exchange and cell counts will be made by flow cytometry after marking with specific fluorescent antibodies (Luminex) and measured as a percentage.
Cycle 5, Group A : T8 DR+ lymphocytes BEFORE single plasma exchange | Day 0, Hour 0
  5 mL of blood will be collected in an EDTA tube BEFORE single plasma exchange and cell counts will be made by flow cytometry after marking with specific fluorescent antibodies (Luminex) and measured as a percentage.
Cycle 5, Group A : B lymphocytes BEFORE single plasma exchange | Day 0, Hour 0
  5 mL of blood will be collected in an EDTA tube BEFORE single plasma exchange and cell counts will be made by flow cytometry after marking with specific fluorescent antibodies (Luminex) and measured as a percentage.
Cycle 5, Group A : CD45RA+CCR7+ cells BEFORE single plasma exchange | Day 0, Hour 0
  5 mL of blood will be collected in an EDTA tube BEFORE single plasma exchange and cell counts will be made by flow cytometry after marking with specific fluorescent antibodies (Luminex) and measured as a percentage.
Cycle 5, Group A : CD45RA-CCR7+ cells BEFORE single plasma exchange | Day 0, Hour 0
  5 mL of blood will be collected in an EDTA tube BEFORE single plasma exchange and cell counts will be made by flow cytometry after marking with specific fluorescent antibodies (Luminex) and measured as a percentage.
Cycle 5, Group A : CD45RA-CCR7- cells BEFORE single plasma exchange | Day 0, Hour 0
  5 mL of blood will be collected in an EDTA tube BEFORE single plasma exchange and cell counts will be made by flow cytometry after marking with specific fluorescent antibodies (Luminex) and measured as a percentage.
Cycle 5, Group A : CCR6-CXCR3- cells BEFORE single plasma exchange | Day 0, Hour 0
  5 mL of blood will be collected in an EDTA tube BEFORE single plasma exchange and cell counts will be made by flow cytometry after marking with specific fluorescent antibodies (Luminex) and measured as a percentage.
Cycle 5, Group A : T4 lymphocytes AFTER single plasma exchange | Day 0, Hour 3
  5 mL of blood will be collected in an EDTA tube AFTER single plasma exchange and cell counts will be made by flow cytometry after marking with specific fluorescent antibodies (Luminex) and measured as a percentage.
Cycle 5, Group A : T4 DR+ lymphocytes AFTER single plasma exchange | Day 0, Hour 3
  5 mL of blood will be collected in an EDTA tube AFTER single plasma exchange and cell counts will be made by flow cytometry after marking with specific fluorescent antibodies (Luminex) and measured as a percentage.
Cycle 5, Group A : T8 lymphocytes AFTER single plasma exchange | Day 0, Hour 3
  5 mL of blood will be collected in an EDTA tube AFTER single plasma exchange and cell counts will be made by flow cytometry after marking with specific fluorescent antibodies (Luminex) and measured as a percentage.
Cycle 5, Group A : T8 DR+ lymphocytes AFTER single plasma exchange | Day 0, Hour 3
  5 mL of blood will be collected in an EDTA tube AFTER single plasma exchange and cell counts will be made by flow cytometry after marking with specific fluorescent antibodies (Luminex) and measured as a percentage.
Cycle 5, Group A : B lymphocytes AFTER single plasma exchange | Day 0, Hour 3
  5 mL of blood will be collected in an EDTA tube AFTER single plasma exchange and cell counts will be made by flow cytometry after marking with specific fluorescent antibodies (Luminex) and measured as a percentage.
Cycle 5, Group A : CD45RA+CCR7+ cells AFTER single plasma exchange | Day 0, Hour 3
  5 mL of blood will be collected in an EDTA tube AFTER single plasma exchange and cell counts will be made by flow cytometry after marking with specific fluorescent antibodies (Luminex) and measured as a percentage.
Cycle 5, Group A : CD45RA-CCR7+ cells AFTER single plasma exchange | Day 0, Hour 3
  5 mL of blood will be collected in an EDTA tube AFTER single plasma exchange and cell counts will be made by flow cytometry after marking with specific fluorescent antibodies (Luminex) and measured as a percentage.
Cycle 5, Group A : CD45RA-CCR7- cells AFTER single plasma exchange | Day 0, Hour 3
  5 mL of blood will be collected in an EDTA tube AFTER single plasma exchange and cell counts will be made by flow cytometry after marking with specific fluorescent antibodies (Luminex) and measured as a percentage.
Cycle 5, Group A : CCR6-CXCR3- cells AFTER single plasma exchange | Day 0, Hour 3
  5 mL of blood will be collected in an EDTA tube AFTER single plasma exchange and cell counts will be made by flow cytometry after marking with specific fluorescent antibodies (Luminex) and measured as a percentage.
Cycle 5, Group A : T4 lymphocytes 7-10 days AFTER single plasma exchange | Day 7-10
  5 mL of blood will be collected in an EDTA tube AFTER single plasma exchange and cell counts will be made by flow cytometry after marking with specific fluorescent antibodies (Luminex) and measured as a percentage.
Cycle 5, Group A : T4 DR+ lymphocytes 7-10 days AFTER single plasma exchange | Day 7-10
  5 mL of blood will be collected in an EDTA tube AFTER single plasma exchange and cell counts will be made by flow cytometry after marking with specific fluorescent antibodies (Luminex) and measured as a percentage.
Cycle 5, Group A : T8 lymphocytes 7-10 days AFTER single plasma exchange | Day 7-10
  5 mL of blood will be collected in an EDTA tube AFTER single plasma exchange and cell counts will be made by flow cytometry after marking with specific fluorescent antibodies (Luminex) and measured as a percentage.
Cycle 5, Group A : T8 DR+ lymphocytes 7-10 days AFTER single plasma exchange | Day 7-10
  5 mL of blood will be collected in an EDTA tube AFTER single plasma exchange and cell counts will be made by flow cytometry after marking with specific fluorescent antibodies (Luminex) and measured as a percentage.
Cycle 5, Group A : B lymphocytes 7-10 days AFTER single plasma exchange | Day 7-10
  5 mL of blood will be collected in an EDTA tube AFTER single plasma exchange and cell counts will be made by flow cytometry after marking with specific fluorescent antibodies (Luminex) and measured as a percentage.
Cycle 5, Group A : CD45RA+CCR7+ cells 7-10 days AFTER single plasma exchange | Day 7-10
  5 mL of blood will be collected in an EDTA tube AFTER single plasma exchange and cell counts will be made by flow cytometry after marking with specific fluorescent antibodies (Luminex) and measured as a percentage.
Cycle 5, Group A : CD45RA-CCR7+ cells 7-10 days AFTER single plasma exchange | Day 7-10
  5 mL of blood will be collected in an EDTA tube AFTER single plasma exchange and cell counts will be made by flow cytometry after marking with specific fluorescent antibodies (Luminex) and measured as a percentage.
Cycle 5, Group A : CD45RA-CCR7- cells 7-10 days AFTER single plasma exchange | Day 7-10
  5 mL of blood will be collected in an EDTA tube AFTER single plasma exchange and cell counts will be made by flow cytometry after marking with specific fluorescent antibodies (Luminex) and measured as a percentage.
Cycle 5, Group A : CCR6-CXCR3- cells 7-10 days AFTER single plasma exchange | Day 7-10
  5 mL of blood will be collected in an EDTA tube AFTER single plasma exchange and cell counts will be made by flow cytometry after marking with specific fluorescent antibodies (Luminex) and measured as a percentage.
Cycle 5, Group B : T4 lymphocytes BEFORE double filtration plasmapheresis | Day 0, Hour 0
  5 mL of blood will be collected in an EDTA tube BEFORE double filtration plasmapheresis and cell counts will be made by flow cytometry after marking with specific fluorescent antibodies (Luminex) and measured as a percentage.
Cycle 5, Group B : T4 DR+ lymphocytes BEFORE double filtration plasmapheresis | Day 0, Hour 0
  5 mL of blood will be collected in an EDTA tube BEFORE double filtration plasmapheresis and cell counts will be made by flow cytometry after marking with specific fluorescent antibodies (Luminex) and measured as a percentage.
Cycle 5, Group B : T8 lymphocytes BEFORE double filtration plasmapheresis | Day 0, Hour 0
  5 mL of blood will be collected in an EDTA tube BEFORE double filtration plasmapheresis and cell counts will be made by flow cytometry after marking with specific fluorescent antibodies (Luminex) and measured as a percentage.
Cycle 5, Group B : T8 DR+ lymphocytes BEFORE double filtration plasmapheresis | Day 0, Hour 0
  5 mL of blood will be collected in an EDTA tube BEFORE double filtration plasmapheresis and cell counts will be made by flow cytometry after marking with specific fluorescent antibodies (Luminex) and measured as a percentage.
Cycle 5, Group B : B lymphocytes BEFORE double filtration plasmapheresis | Day 0, Hour 0
  5 mL of blood will be collected in an EDTA tube BEFORE double filtration plasmapheresis and cell counts will be made by flow cytometry after marking with specific fluorescent antibodies (Luminex) and measured as a percentage.
Cycle 5, Group B : CD45RA+CCR7+ cells BEFORE double filtration plasmapheresis | Day 0, Hour 0
  5 mL of blood will be collected in an EDTA tube BEFORE double filtration plasmapheresis and cell counts will be made by flow cytometry after marking with specific fluorescent antibodies (Luminex) and measured as a percentage.
Cycle 5, Group B : CD45RA-CCR7+ cells BEFORE double filtration plasmapheresis | Day 0, Hour 0
  5 mL of blood will be collected in an EDTA tube BEFORE double filtration plasmapheresis and cell counts will be made by flow cytometry after marking with specific fluorescent antibodies (Luminex) and measured as a percentage.
Cycle 5, Group B : CD45RA-CCR7- cells BEFORE double filtration plasmapheresis | Day 0, Hour 0
  5 mL of blood will be collected in an EDTA tube BEFORE double filtration plasmapheresis and cell counts will be made by flow cytometry after marking with specific fluorescent antibodies (Luminex) and measured as a percentage.
Cycle 5, Group B : CCR6-CXCR3- cells BEFORE double filtration plasmapheresis | Day 0, Hour 0
  5 mL of blood will be collected in an EDTA tube BEFORE double filtration plasmapheresis and cell counts will be made by flow cytometry after marking with specific fluorescent antibodies (Luminex) and measured as a percentage.
Cycle 5, Group B : T4 lymphocytes AFTER double filtration plasmapheresis | Day 0, Hour 3
  5 mL of blood will be collected in an EDTA tube AFTER double filtration plasmapheresis and cell counts will be made by flow cytometry after marking with specific fluorescent antibodies (Luminex) and measured as a percentage.
Cycle 5, Group B : T4 DR+ lymphocytes AFTER double filtration plasmapheresis | Day 0, Hour 3
  5 mL of blood will be collected in an EDTA tube AFTER double filtration plasmapheresis and cell counts will be made by flow cytometry after marking with specific fluorescent antibodies (Luminex) and measured as a percentage.
Cycle 5, Group B : T8 lymphocytes AFTER double filtration plasmapheresis | Day 0, Hour 3
  5 mL of blood will be collected in an EDTA tube AFTER double filtration plasmapheresis and cell counts will be made by flow cytometry after marking with specific fluorescent antibodies (Luminex) and measured as a percentage.
Cycle 5, Group B : T8 DR+ lymphocytes AFTER double filtration plasmapheresis | Day 0, Hour 3
  5 mL of blood will be collected in an EDTA tube AFTER double filtration plasmapheresis and cell counts will be made by flow cytometry after marking with specific fluorescent antibodies (Luminex) and measured as a percentage.
Cycle 5, Group B : B lymphocytes AFTER double filtration plasmapheresis | Day 0, Hour 3
  5 mL of blood will be collected in an EDTA tube AFTER double filtration plasmapheresis and cell counts will be made by flow cytometry after marking with specific fluorescent antibodies (Luminex) and measured as a percentage.
Cycle 5, Group B : CD45RA+CCR7+ cells AFTER double filtration plasmapheresis | Day 0, Hour 3
  5 mL of blood will be collected in an EDTA tube AFTER double filtration plasmapheresis and cell counts will be made by flow cytometry after marking with specific fluorescent antibodies (Luminex) and measured as a percentage.
Cycle 5, Group B : CD45RA-CCR7+ cells AFTER double filtration plasmapheresis | Day 0, Hour 3
  5 mL of blood will be collected in an EDTA tube AFTER double filtration plasmapheresis and cell counts will be made by flow cytometry after marking with specific fluorescent antibodies (Luminex) and measured as a percentage.
Cycle 5, Group B : CD45RA-CCR7- cells AFTER double filtration plasmapheresis | Day 0, Hour 3
  5 mL of blood will be collected in an EDTA tube AFTER double filtration plasmapheresis and cell counts will be made by flow cytometry after marking with specific fluorescent antibodies (Luminex) and measured as a percentage.
Cycle 5, Group B : CCR6-CXCR3- cells AFTER double filtration plasmapheresis | Day 0, Hour 3
  5 mL of blood will be collected in an EDTA tube AFTER double filtration plasmapheresis and cell counts will be made by flow cytometry after marking with specific fluorescent antibodies (Luminex) and measured as a percentage.
Cycle 5, Group B : T4 lymphocytes 7-10 days AFTER double filtration plasmapheresis | Day 7-10
  5 mL of blood will be collected in an EDTA tube AFTER double filtration plasmapheresis and cell counts will be made by flow cytometry after marking with specific fluorescent antibodies (Luminex) and measured as a percentage.
Cycle 5, Group B : T4 DR+ lymphocytes 7-10 days AFTER double filtration plasmapheresis | Day 7-10
  5 mL of blood will be collected in an EDTA tube AFTER double filtration plasmapheresis and cell counts will be made by flow cytometry after marking with specific fluorescent antibodies (Luminex) and measured as a percentage.
Cycle 5, Group B : T8 lymphocytes 7-10 days AFTER double filtration plasmapheresis | Day 7-10
  5 mL of blood will be collected in an EDTA tube AFTER double filtration plasmapheresis and cell counts will be made by flow cytometry after marking with specific fluorescent antibodies (Luminex) and measured as a percentage.
Cycle 5, Group B : T8 DR+ lymphocytes 7-10 days AFTER double filtration plasmapheresis | Day 7-10
  5 mL of blood will be collected in an EDTA tube AFTER double filtration plasmapheresis and cell counts will be made by flow cytometry after marking with specific fluorescent antibodies (Luminex) and measured as a percentage.
Cycle 5, Group B : B lymphocytes 7-10 days AFTER double filtration plasmapheresis | Day 7-10
  5 mL of blood will be collected in an EDTA tube AFTER double filtration plasmapheresis and cell counts will be made by flow cytometry after marking with specific fluorescent antibodies (Luminex) and measured as a percentage.
Cycle 5, Group B : CD45RA+CCR7+ cells 7-10 days AFTER double filtration plasmapheresis | Day 7-10
  5 mL of blood will be collected in an EDTA tube AFTER double filtration plasmapheresis and cell counts will be made by flow cytometry after marking with specific fluorescent antibodies (Luminex) and measured as a percentage.
Cycle 5, Group B : CD45RA-CCR7+ cells 7-10 days AFTER double filtration plasmapheresis | Day 7-10
  5 mL of blood will be collected in an EDTA tube AFTER double filtration plasmapheresis and cell counts will be made by flow cytometry after marking with specific fluorescent antibodies (Luminex) and measured as a percentage.
Cycle 5, Group B : CD45RA-CCR7- cells 7-10 days AFTER double filtration plasmapheresis | Day 7-10
  5 mL of blood will be collected in an EDTA tube AFTER double filtration plasmapheresis and cell counts will be made by flow cytometry after marking with specific fluorescent antibodies (Luminex) and measured as a percentage.
Cycle 5, Group B : CCR6-CXCR3- cells 7-10 days AFTER double filtration plasmapheresis | Day 7-10
  5 mL of blood will be collected in an EDTA tube AFTER double filtration plasmapheresis and cell counts will be made by flow cytometry after marking with specific fluorescent antibodies (Luminex) and measured as a percentage.
Cycle 6, Group A : T4 lymphocytes BEFORE double filtration plasmapheresis | Day 0, Hour 0
  5 mL of blood will be collected in an EDTA tube BEFORE double filtration plasmapheresis and cell counts will be made by flow cytometry after marking with specific fluorescent antibodies (Luminex) and measured as a percentage.
Cycle 6, Group A : T4 DR+ lymphocytes BEFORE double filtration plasmapheresis | Day 0, Hour 0
  5 mL of blood will be collected in an EDTA tube BEFORE double filtration plasmapheresis and cell counts will be made by flow cytometry after marking with specific fluorescent antibodies (Luminex) and measured as a percentage.
Cycle 6, Group A : T8 lymphocytes BEFORE double filtration plasmapheresis | Day 0, Hour 0
  5 mL of blood will be collected in an EDTA tube BEFORE double filtration plasmapheresis and cell counts will be made by flow cytometry after marking with specific fluorescent antibodies (Luminex) and measured as a percentage.
Cycle 6, Group A : T8 DR+ lymphocytes BEFORE double filtration plasmapheresis | Day 0, Hour 0
  5 mL of blood will be collected in an EDTA tube BEFORE double filtration plasmapheresis and cell counts will be made by flow cytometry after marking with specific fluorescent antibodies (Luminex) and measured as a percentage.
Cycle 6, Group A : B lymphocytes BEFORE double filtration plasmapheresis | Day 0, Hour 0
  5 mL of blood will be collected in an EDTA tube BEFORE double filtration plasmapheresis and cell counts will be made by flow cytometry after marking with specific fluorescent antibodies (Luminex) and measured as a percentage.
Cycle 6, Group A : CD45RA+CCR7+ cells BEFORE double filtration plasmapheresis | Day 0, Hour 0
  5 mL of blood will be collected in an EDTA tube BEFORE double filtration plasmapheresis and cell counts will be made by flow cytometry after marking with specific fluorescent antibodies (Luminex) and measured as a percentage.
Cycle 6, Group A : CD45RA-CCR7+ cells BEFORE double filtration plasmapheresis | Day 0, Hour 0
  5 mL of blood will be collected in an EDTA tube BEFORE double filtration plasmapheresis and cell counts will be made by flow cytometry after marking with specific fluorescent antibodies (Luminex) and measured as a percentage.
Cycle 6, Group A : CD45RA-CCR7- cells BEFORE double filtration plasmapheresis | Day 0, Hour 0
  5 mL of blood will be collected in an EDTA tube BEFORE double filtration plasmapheresis and cell counts will be made by flow cytometry after marking with specific fluorescent antibodies (Luminex) and measured as a percentage.
Cycle 6, Group A : CCR6-CXCR3- cells BEFORE double filtration plasmapheresis | Day 0, Hour 0
  5 mL of blood will be collected in an EDTA tube BEFORE double filtration plasmapheresis and cell counts will be made by flow cytometry after marking with specific fluorescent antibodies (Luminex) and measured as a percentage.
Cycle 6, Group A : T4 lymphocytes AFTER double filtration plasmapheresis | Day 0, Hour 3
  5 mL of blood will be collected in an EDTA tube AFTER double filtration plasmapheresis and cell counts will be made by flow cytometry after marking with specific fluorescent antibodies (Luminex) and measured as a percentage.
Cycle 6, Group A : T4 DR+ lymphocytes AFTER double filtration plasmapheresis | Day 0, Hour 3
  5 mL of blood will be collected in an EDTA tube AFTER double filtration plasmapheresis and cell counts will be made by flow cytometry after marking with specific fluorescent antibodies (Luminex) and measured as a percentage.
Cycle 6, Group A : T8 lymphocytes AFTER double filtration plasmapheresis | Day 0, Hour 3
  5 mL of blood will be collected in an EDTA tube AFTER double filtration plasmapheresis and cell counts will be made by flow cytometry after marking with specific fluorescent antibodies (Luminex) and measured as a percentage.
Cycle 6, Group A : T8 DR+ lymphocytes AFTER double filtration plasmapheresis | Day 0, Hour 3
  5 mL of blood will be collected in an EDTA tube AFTER double filtration plasmapheresis and cell counts will be made by flow cytometry after marking with specific fluorescent antibodies (Luminex) and measured as a percentage.
Cycle 6, Group A : B lymphocytes AFTER double filtration plasmapheresis | Day 0, Hour 3
  5 mL of blood will be collected in an EDTA tube AFTER double filtration plasmapheresis and cell counts will be made by flow cytometry after marking with specific fluorescent antibodies (Luminex) and measured as a percentage.
Cycle 6, Group A : CD45RA+CCR7+ cells AFTER double filtration plasmapheresis | Day 0, Hour 3
  5 mL of blood will be collected in an EDTA tube AFTER double filtration plasmapheresis and cell counts will be made by flow cytometry after marking with specific fluorescent antibodies (Luminex) and measured as a percentage.
Cycle 6, Group A : CD45RA-CCR7+ cells AFTER double filtration plasmapheresis | Day 0, Hour 3
  5 mL of blood will be collected in an EDTA tube AFTER double filtration plasmapheresis and cell counts will be made by flow cytometry after marking with specific fluorescent antibodies (Luminex) and measured as a percentage.
Cycle 6, Group A : CD45RA-CCR7- cells AFTER double filtration plasmapheresis | Day 0, Hour 3
  5 mL of blood will be collected in an EDTA tube AFTER double filtration plasmapheresis and cell counts will be made by flow cytometry after marking with specific fluorescent antibodies (Luminex) and measured as a percentage.
Cycle 6, Group A : CCR6-CXCR3- cells AFTER double filtration plasmapheresis | Day 0, Hour 3
  5 mL of blood will be collected in an EDTA tube AFTER double filtration plasmapheresis and cell counts will be made by flow cytometry after marking with specific fluorescent antibodies (Luminex) and measured as a percentage.
Cycle 6, Group A : T4 lymphocytes 7-10 days AFTER double filtration plasmapheresis | Day 7-10
  5 mL of blood will be collected in an EDTA tube AFTER double filtration plasmapheresis and cell counts will be made by flow cytometry after marking with specific fluorescent antibodies (Luminex) and measured as a percentage.
Cycle 6, Group A : T4 DR+ lymphocytes 7-10 days AFTER double filtration plasmapheresis | Day 7-10
  5 mL of blood will be collected in an EDTA tube AFTER double filtration plasmapheresis and cell counts will be made by flow cytometry after marking with specific fluorescent antibodies (Luminex) and measured as a percentage.
Cycle 6, Group A : T8 lymphocytes 7-10 days AFTER double filtration plasmapheresis | Day 7-10
  5 mL of blood will be collected in an EDTA tube AFTER double filtration plasmapheresis and cell counts will be made by flow cytometry after marking with specific fluorescent antibodies (Luminex) and measured as a percentage.
Cycle 6, Group A : T8 DR+ lymphocytes 7-10 days AFTER double filtration plasmapheresis | Day 7-10
  5 mL of blood will be collected in an EDTA tube AFTER double filtration plasmapheresis and cell counts will be made by flow cytometry after marking with specific fluorescent antibodies (Luminex) and measured as a percentage.
Cycle 6, Group A : B lymphocytes 7-10 days AFTER double filtration plasmapheresis | Day 7-10
  5 mL of blood will be collected in an EDTA tube AFTER double filtration plasmapheresis and cell counts will be made by flow cytometry after marking with specific fluorescent antibodies (Luminex) and measured as a percentage.
Cycle 6, Group A : CD45RA+CCR7+ cells 7-10 days AFTER double filtration plasmapheresis | Day 7-10
  5 mL of blood will be collected in an EDTA tube AFTER double filtration plasmapheresis and cell counts will be made by flow cytometry after marking with specific fluorescent antibodies (Luminex) and measured as a percentage.
Cycle 6, Group A : CD45RA-CCR7+ cells 7-10 days AFTER double filtration plasmapheresis | Day 7-10
  5 mL of blood will be collected in an EDTA tube AFTER double filtration plasmapheresis and cell counts will be made by flow cytometry after marking with specific fluorescent antibodies (Luminex) and measured as a percentage.
Cycle 6, Group A : CD45RA-CCR7- cells 7-10 days AFTER double filtration plasmapheresis | Day 7-10
  5 mL of blood will be collected in an EDTA tube AFTER double filtration plasmapheresis and cell counts will be made by flow cytometry after marking with specific fluorescent antibodies (Luminex) and measured as a percentage.
Cycle 6, Group A : CCR6-CXCR3- cells 7-10 days AFTER double filtration plasmapheresis | Day 7-10
  5 mL of blood will be collected in an EDTA tube AFTER double filtration plasmapheresis and cell counts will be made by flow cytometry after marking with specific fluorescent antibodies (Luminex) and measured as a percentage.
Cycle 6, Group B : T4 lymphocytes BEFORE single plasma exchange | Day 0, H0
  5 mL of blood will be collected in an EDTA tube BEFORE single plasma exchange and cell counts will be made by flow cytometry after marking with specific fluorescent antibodies (Luminex) and measured as a percentage.
Cycle 6, Group B : T4 DR+ lymphocytes BEFORE single plasma exchange | Day 0, H0
  5 mL of blood will be collected in an EDTA tube BEFORE single plasma exchange and cell counts will be made by flow cytometry after marking with specific fluorescent antibodies (Luminex) and measured as a percentage.
Cycle 6, Group B : T8 lymphocytes BEFORE single plasma exchange | Day 0, H0
  5 mL of blood will be collected in an EDTA tube BEFORE single plasma exchange and cell counts will be made by flow cytometry after marking with specific fluorescent antibodies (Luminex) and measured as a percentage.
Cycle 6, Group B : T8 DR+ lymphocytes BEFORE single plasma exchange | Day 0, H0
  5 mL of blood will be collected in an EDTA tube BEFORE single plasma exchange and cell counts will be made by flow cytometry after marking with specific fluorescent antibodies (Luminex) and measured as a percentage.
Cycle 6, Group B : B lymphocytes BEFORE single plasma exchange | Day 0, H0
  5 mL of blood will be collected in an EDTA tube BEFORE single plasma exchange and cell counts will be made by flow cytometry after marking with specific fluorescent antibodies (Luminex) and measured as a percentage.
Cycle 6, Group B : CD45RA+CCR7+ cells BEFORE single plasma exchange | Day 0, H0
  5 mL of blood will be collected in an EDTA tube BEFORE single plasma exchange and cell counts will be made by flow cytometry after marking with specific fluorescent antibodies (Luminex) and measured as a percentage.
Cycle 6, Group B : CD45RA-CCR7+ cells BEFORE single plasma exchange | Day 0, H0
  5 mL of blood will be collected in an EDTA tube BEFORE single plasma exchange and cell counts will be made by flow cytometry after marking with specific fluorescent antibodies (Luminex) and measured as a percentage.
Cycle 6, Group B : CD45RA-CCR7- cells BEFORE single plasma exchange | Day 0, H0
  5 mL of blood will be collected in an EDTA tube BEFORE single plasma exchange and cell counts will be made by flow cytometry after marking with specific fluorescent antibodies (Luminex) and measured as a percentage.
Cycle 6, Group B : CCR6-CXCR3- cells BEFORE single plasma exchange | Day 0, H0
  5 mL of blood will be collected in an EDTA tube BEFORE single plasma exchange and cell counts will be made by flow cytometry after marking with specific fluorescent antibodies (Luminex) and measured as a percentage.
Cycle 6, Group B : T4 lymphocytes AFTER single plasma exchange | Day 0, H3
  5 mL of blood will be collected in an EDTA tube AFTER single plasma exchange and cell counts will be made by flow cytometry after marking with specific fluorescent antibodies (Luminex) and measured as a percentage.
Cycle 6, Group B : T4 DR+ lymphocytes AFTER single plasma exchange | Day 0, H3
  5 mL of blood will be collected in an EDTA tube AFTER single plasma exchange and cell counts will be made by flow cytometry after marking with specific fluorescent antibodies (Luminex) and measured as a percentage.
Cycle 6, Group B : T8 lymphocytes AFTER single plasma exchange | Day 0, H3
  5 mL of blood will be collected in an EDTA tube AFTER single plasma exchange and cell counts will be made by flow cytometry after marking with specific fluorescent antibodies (Luminex) and measured as a percentage.
Cycle 6, Group B : T8 DR+ lymphocytes AFTER single plasma exchange | Day 0, H3
  5 mL of blood will be collected in an EDTA tube AFTER single plasma exchange and cell counts will be made by flow cytometry after marking with specific fluorescent antibodies (Luminex) and measured as a percentage.
Cycle 6, Group B : B lymphocytes AFTER single plasma exchange | Day 0, H3
  5 mL of blood will be collected in an EDTA tube AFTER single plasma exchange and cell counts will be made by flow cytometry after marking with specific fluorescent antibodies (Luminex) and measured as a percentage.
Cycle 6, Group B : CD45RA+CCR7+ cells AFTER single plasma exchange | Day 0, H3
  5 mL of blood will be collected in an EDTA tube AFTER single plasma exchange and cell counts will be made by flow cytometry after marking with specific fluorescent antibodies (Luminex) and measured as a percentage.
Cycle 6, Group B : CD45RA-CCR7+ cells AFTER single plasma exchange | Day 0, H3
  5 mL of blood will be collected in an EDTA tube AFTER single plasma exchange and cell counts will be made by flow cytometry after marking with specific fluorescent antibodies (Luminex) and measured as a percentage.
Cycle 6, Group B : CD45RA-CCR7- cells AFTER single plasma exchange | Day 0, H3
  5 mL of blood will be collected in an EDTA tube AFTER single plasma exchange and cell counts will be made by flow cytometry after marking with specific fluorescent antibodies (Luminex) and measured as a percentage.
Cycle 6, Group B : CCR6-CXCR3- cells AFTER single plasma exchange | Day 0, H3
  5 mL of blood will be collected in an EDTA tube AFTER single plasma exchange and cell counts will be made by flow cytometry after marking with specific fluorescent antibodies (Luminex) and measured as a percentage.
Cycle 6, Group B : T4 lymphocytes 7-10 days AFTER single plasma exchange | Day 7-10
  5 mL of blood will be collected in an EDTA tube AFTER single plasma exchange and cell counts will be made by flow cytometry after marking with specific fluorescent antibodies (Luminex) and measured as a percentage.
Cycle 6, Group B : T4 DR+ lymphocytes 7-10 days AFTER single plasma exchange | Day 7-10
  5 mL of blood will be collected in an EDTA tube AFTER single plasma exchange and cell counts will be made by flow cytometry after marking with specific fluorescent antibodies (Luminex) and measured as a percentage.
Cycle 6, Group B : T8 lymphocytes 7-10 days AFTER single plasma exchange | Day 7-10
  5 mL of blood will be collected in an EDTA tube AFTER single plasma exchange and cell counts will be made by flow cytometry after marking with specific fluorescent antibodies (Luminex) and measured as a percentage.
Cycle 6, Group B : T8 DR+ lymphocytes 7-10 days AFTER single plasma exchange | Day 7-10
  5 mL of blood will be collected in an EDTA tube AFTER single plasma exchange and cell counts will be made by flow cytometry after marking with specific fluorescent antibodies (Luminex) and measured as a percentage.
Cycle 6, Group B : B lymphocytes 7-10 days AFTER single plasma exchange | Day 7-10
  5 mL of blood will be collected in an EDTA tube AFTER single plasma exchange and cell counts will be made by flow cytometry after marking with specific fluorescent antibodies (Luminex) and measured as a percentage.
Cycle 6, Group B : CD45RA+CCR7+ cells 7-10 days AFTER single plasma exchange | Day 7-10
  5 mL of blood will be collected in an EDTA tube AFTER single plasma exchange and cell counts will be made by flow cytometry after marking with specific fluorescent antibodies (Luminex) and measured as a percentage.
Cycle 6, Group B : CD45RA-CCR7+ cells 7-10 days AFTER single plasma exchange | Day 7-10
  5 mL of blood will be collected in an EDTA tube AFTER single plasma exchange and cell counts will be made by flow cytometry after marking with specific fluorescent antibodies (Luminex) and measured as a percentage.
Cycle 6, Group B : CD45RA-CCR7- cells 7-10 days AFTER single plasma exchange | Day 7-10
  5 mL of blood will be collected in an EDTA tube AFTER single plasma exchange and cell counts will be made by flow cytometry after marking with specific fluorescent antibodies (Luminex) and measured as a percentage.
Cycle 6, Group B : CCR6-CXCR3- cells 7-10 days AFTER single plasma exchange | Day 7-10
  5 mL of blood will be collected in an EDTA tube AFTER single plasma exchange and cell counts will be made by flow cytometry after marking with specific fluorescent antibodies (Luminex) and measured as a percentage.

OTHER OUTCOMES:
Group A, Cycle 1 : Link between variations in lymphocyte sub-populations and the clinical evolution . | Day 7-10 after the end of Cycle 1 (each cycle lasts 3 hours)
  All the above primary and secondary outcome measures will be compared with clinical information in the patient file in order to determine a link between these variations at the end of each treatment cycle.
Group B, Cycle 1 : Link between variations in lymphocyte sub-populations and the clinical evolution . | Day 7-10 after the end of Cycle 1 (each cycle lasts 3 hours)
  All the above primary and secondary outcome measures will be compared with clinical information in the patient file in order to determine a link between these variations at the end of each treatment cycle.
Group A, Cycle 2 : Link between variations in lymphocyte sub-populations and the clinical evolution . | Day 7-10 after the end of Cycle 2 (each cycle lasts 3 hours)
  All the above primary and secondary outcome measures will be compared with clinical information in the patient file in order to determine a link between these variations at the end of each treatment cycle.
Group B, Cycle 2 : Link between variations in lymphocyte sub-populations and the clinical evolution . | Day 7-10 after the end of Cycle 2 (each cycle lasts 3 hours)
  All the above primary and secondary outcome measures will be compared with clinical information in the patient file in order to determine a link between these variations at the end of each treatment cycle.
Group A, Cycle 3 : Link between variations in lymphocyte sub-populations and the clinical evolution . | Day 7-10 after the end of Cycle 3 (each cycle lasts 3 hours)
  All the above primary and secondary outcome measures will be compared with clinical information in the patient file in order to determine a link between these variations at the end of each treatment cycle.
Group B, Cycle 3 : Link between variations in lymphocyte sub-populations and the clinical evolution . | Day 7-10 after the end of Cycle 3 (each cycle lasts 3 hours)
  All the above primary and secondary outcome measures will be compared with clinical information in the patient file in order to determine a link between these variations at the end of each treatment cycle.
Group A, Cycle 4 : Link between variations in lymphocyte sub-populations and the clinical evolution . | Day 7-10 after the end of Cycle 4 (each cycle lasts 3 hours)
  All the above primary and secondary outcome measures will be compared with clinical information in the patient file in order to determine a link between these variations at the end of each treatment cycle.
Group B, Cycle 4 : Link between variations in lymphocyte sub-populations and the clinical evolution . | Day 7-10 after the end of Cycle 4 (each cycle lasts 3 hours)
  All the above primary and secondary outcome measures will be compared with clinical information in the patient file in order to determine a link between these variations at the end of each treatment cycle.
Group A, Cycle 5 : Link between variations in lymphocyte sub-populations and the clinical evolution . | Day 7-10 after the end of Cycle 5 (each cycle lasts 3 hours)
  All the above primary and secondary outcome measures will be compared with clinical information in the patient file in order to determine a link between these variations at the end of each treatment cycle.
Group B, Cycle 5 : Link between variations in lymphocyte sub-populations and the clinical evolution . | Day 7-10 after the end of Cycle 5 (each cycle lasts 3 hours)
  All the above primary and secondary outcome measures will be compared with clinical information in the patient file in order to determine a link between these variations at the end of each treatment cycle.
Group A, Cycle 6 : Link between variations in lymphocyte sub-populations and the clinical evolution . | Day 7-10 after the end of Cycle 6 (each cycle lasts 3 hours)
  All the above primary and secondary outcome measures will be compared with clinical information in the patient file in order to determine a link between these variations at the end of each treatment cycle.
Group B, Cycle 6 : Link between variations in lymphocyte sub-populations and the clinical evolution . | Day 7-10 after the end of Cycle 6 (each cycle lasts 3 hours)
  All the above primary and secondary outcome measures will be compared with clinical information in the patient file in order to determine a link between these variations at the end of each treatment cycle.
Group A, Cycle 1 : Cost of single plasma exchange to the health institution. | Day 7-10 after the end of Cycle 1 (each cycle lasts 3 hours)
  The cost of each cycle will be recorded in Euros in the electronic clinical research file and the average amount will be calculated from this information at the end of 6 cycles.
Group B, Cycle 1 : Cost of double filtration plasmapheresis to the health institution. | Day 7-10 after the end of Cycle 1 (each cycle lasts 3 hours)
  The cost of each cycle will be recorded in Euros in the electronic clinical research file and the average amount will be calculated from this information at the end of 6 cycles.
Group A, Cycle 2 : Cost of double filtration plasmapheresis to the health institution. | Day 7-10 after the end of Cycle 2 (each cycle lasts 3 hours)
  The cost of each cycle will be recorded in Euros in the electronic clinical research file and the average amount will be calculated from this information at the end of 6 cycles.
Group B, Cycle 2 : Cost of single plasma exchange to the health institution. | Day 7-10 after the end of Cycle 2 (each cycle lasts 3 hours)
  The cost of each cycle will be recorded in Euros in the electronic clinical research file and the average amount will be calculated from this information at the end of 6 cycles.
Group A, Cycle 3 : Cost of single plasma exchange to the health institution. | Day 7-10 after the end of Cycle 3 (each cycle lasts 3 hours)
  The cost of each cycle will be recorded in Euros in the electronic clinical research file and the average amount will be calculated from this information at the end of 6 cycles.
Group B, Cycle 3 : Cost of double filtration plasmapheresis to the health institution. | Day 7-10 after the end of Cycle 3 (each cycle lasts 3 hours)
  The cost of each cycle will be recorded in Euros in the electronic clinical research file and the average amount will be calculated from this information at the end of 6 cycles.
Group A, Cycle 4 : Cost of double filtration plasmapheresis to the health institution. | Day 7-10 after the end of Cycle 4 (each cycle lasts 3 hours)
  The cost of each cycle will be recorded in Euros in the electronic clinical research file and the average amount will be calculated from this information at the end of 6 cycles.
Group B, Cycle 4 : Cost of single plasma exchange to the health institution. | Day 7-10 after the end of Cycle 4 (each cycle lasts 3 hours)
  The cost of each cycle will be recorded in Euros in the electronic clinical research file and the average amount will be calculated from this information at the end of 6 cycles.
Group A, Cycle 5 : Cost of single plasma exchange to the health institution. | Day 7-10 after the end of Cycle 5 (each cycle lasts 3 hours)
  The cost of each cycle will be recorded in Euros in the electronic clinical research file and the average amount will be calculated from this information at the end of 6 cycles.
Group B, Cycle 5 : Cost of double filtration to the health institution. | Day 7-10 after the end of Cycle 5 (each cycle lasts 3 hours)
  The cost of each cycle will be recorded in Euros in the electronic clinical research file and the average amount will be calculated from this information at the end of 6 cycles.
Group A, Cycle 6 : Cost of double filtration to the health institution. | Day 7-10 after the end of Cycle 6 (each cycle lasts 3 hours)
  The cost of each cycle will be recorded in Euros in the electronic clinical research file and the average amount will be calculated from this information at the end of 6 cycles.
Group B, Cycle 6 : Cost of double filtration to the health institution. | Day 7-10 after the end of Cycle 6 (each cycle lasts 3 hours)
  The cost of each cycle will be recorded in Euros in the electronic clinical research file and the average amount will be calculated from this information at the end of 6 cycles.
Constitution of a biological resource centre using the blood samples taken in view of future research, especially immunological phenotyping. | Day 0, Hour 0
  After all the above analyses, the unused aliquots from the samples taken (bottom of tubes) will be conserved and indexed.
Constitution of a biological resource centre using the blood samples taken in view of future research, especially immunological phenotyping. | Day 0, Hour 3
  After all the above analyses, the unused aliquots from the samples taken (bottom of tubes) will be conserved and indexed.
Constitution of a biological resource centre using the blood samples taken in view of future research, especially immunological phenotyping. | Day 7-10
  After all the above analyses, the unused aliquots from the samples taken (bottom of tubes) will be conserved and indexed.
Compare lymphocyte phenotype between patients with PIDC and control subjects. | Day 0
  Significant difference in Th1/Th2 ratio between PIDC patients and control subjects.

CONTACTS AND LOCATIONS:
Locations (1):
- Olivier MORANNE, Nîmes, France

REFERENCES:
- [Background] Moranne O, Ion IM, Cezar R, Messikh Z, Prelipcean C, Chkair S, Thouvenot E, Tran TA, Corbeau P, Chevallier T. Protocol of comparison of the effects of single plasma exchange and double filtration plasmapheresis on peripheral lymphocyte phenotypes in patients with Chronic Inflammatory Demyelinating Polyradiculoneuropathy: a monocentric prospective study with single-case experimental design. BMC Neurol. 2022 Aug 5;22(1):293. doi: 10.1186/s12883-022-02816-w. PMID 35931957